

# CTN-0051

# Extended-Release Naltrexone vs. Buprenorphine for Opioid Treatment (X:BOT)

**Statistical Analysis Plan (SAP)** 

Version 3.0

April 27, 2017

# **Table of Contents**

| LIST OF ABBI | REVIATIONS | 6 |
|---|---|---|
| LIST OF ABBI | REVIATIONS (cont.) | 7 |
| 1.0 INTRO | DDUCTION | 8 |
| | y Objective | |
| | y Design | |
| | tment Initiation | |
| | Study Data Analysis Modification | |
| | base Sources | |
| | domizationy Population | |
| | Inclusion Criteria | |
| | Exclusion Criteria | |
| | OMES | |
| | ary Outcome | |
| | ondary Outcomes | |
| | RAL CONSIDERATIONS | |
| | ninations | |
| 3.2 Stud | y Modification for Differential Treatment Initiation | 16 |
| | ple Size and Power Calculations | |
| | im Analysis | |
| | vareysis Populations | |
| | ibutional Assumption Tests | |
| 4.0 ANALY | YSES OF DEMOGRAPHIC AND BASELINE DATA | .21 |
| 5.0 STATI | STICAL ANALYSES | .22 |
| 5.1 Timir | ng of Randomization Definitions | 22 |
| 5.2 Diffe | rential Treatment Initiation for Early Randomizers Assessment | 22 |
| 5.2.1 I | Induction Status Determination | 22 |
| 5.2.2 I | Induction Status Analysis | 22 |
| 5.3 Prim | ary Outcome | 22 |
| 5.3.1 F | Primary Outcome Criteria | 23 |
| 5.3.3 I | Primary Outcome Analysis Methods | 25 |
| | ondary Analyses of Primary Outcome Measure | |
| | ondary Outcomes | |
| | Induction Success | |
| 5.5.2 | Opioid Abstinence | 28 |
| | Cigarette Smoking | |
| 5.5.4 | Opioid Craving | 28 |
| 5.5.5 | Subacute Withdrawal Symptoms | 28 |
| 5.5.6 I | Drug Use Problems | 28 |
| 5.5.7 I | HIV Risk Behavior as Assessed by the RAB | 29 |
| 5.5.8 | Cognitive Function | 29 |

| 5.6 Minority/Gender Analyses | |
|---|---|
| 6.0 MISSING DATA | 30 |
| 7.0 SAFETY ANALYSES | |
| 7.1 Physical Examination | |
| 7.2 Concise Health Risk Tracking-Self Report (CHRT-SR) | |
| 7.3 The Hamilton Depression Scale (17 item) (HAM-D) | |
| 7.4.1 Adverse Events (AEs) and Serious Adverse Events (SAEs) | |
| 7.5 Injection Site Examination | |
| 8.0 REFERENCES | |
| Listing of Tables and Figures | |
| Table 1: Protocol Secondary Outcomes and Hypotheses | 13 |
| Table 2: Detectable Alternatives and Power for 2-tailed 5% level logrank test without of | |
| Null distribution has a 40% 6 month success rate, N1=N2=200 | |
| Table 3: CTN-0051 Protocol Calendar | |
| Table 4: Determination of the Start of the Clinical Qualifying Event | 25 |
| Listing of Appendix A Tables and Figures | |
| Figure 1: Consort Diagram | 35 |
| Figure 2: Randomization Status by CTP | |
| Figure 3: Overall Expected vs. Actual Randomizations | |
| Figure 4A: Early Randomizers Actual Randomizations | |
| Figure 5B: Late Randomizers Actual Randomizations | |
| Table 1: Summary of Consents, Eligible Screens and Randomizations by CTP | |
| Table 2: Summary of Screen Failures by CTP | |
| Table 3: Summary of the Timing of Randomization by CTP | |
| Table 4: Summary of Participant Study Disposition by Treatment Arm | |
| Table 5: Randomization by CTP and Stratification Factor | |
| Table 5a: Randomization by CTP and Stratification Factor for Early Randomizers | |
| Table 5b: Randomization by CTP and Stratification Factor for Late Randomizers | |
| Table 6: Summary of Study Medication Induction by Treatment Arm | |
| Table 7: Summary of Induction Status for the Groups of Interest | |
| Table 8: Summary of Early Medication Terminations* by Treatment Arm | |
| Table 9: Summary of Baseline Characteristics by Treatment Arm | |
| Table 10: Summary of Baseline Moderators by Treatment Arm | |
| rable 10. Canimary of Eaconite Moderators by Treatment 74111 | |

| Table 12: Summary of Vivitrol Injections and Injection Intervals by CTP | |
|---|---|
| Table 13: Summary of BUP-NX Prescribed Daily Dose by CTP | 57 |
| Figure 6: Participant-level Prescribed Daily Dose of Buprenorphine | |
| Table 14: Availability of Primary Outcome by Treatment Arm (Day 21 – Day 167*) | 59 |
| Table 15: Summary of Primary Outcome (Relapse) by Treatment Arm | 60 |
| Figure 5A: TLFB and UDS for Day 0 to Day 21Figure 5A: UDS for Day 0 to Day 21- | |
| Treatment=BUP-NX | |
| Figure 5B: UDS for Day 0 to Day 21- Treatment=XR-NTX | |
| Figure 5C: TLFB for Day 0 to Day 21- Treatment=BUP-NX | |
| Figure 5D: TLFB for Day 0 to Day 21- Treatment=XR-NTX | |
| Figure 6: Kaplan-Meier Plots of Time to Relapse by Treatment Arm | |
| Table 16: Summary of Primary Outcome (Time to Relapse <sup>1</sup> ) for Groups of Interest | 63 |
| Figure 7: Kaplan-Meier Plots of Time to Relapse by Randomization Timing Status and Treatment Arm | 64 |
| Figure 8: Kaplan-Meier Plots of Time to Relapse by Opioid Severity Level and Treatment | Arm65 |
| Figure 9: Kaplan-Meier Plots of Time to Relapse by Randomization Timing, Opioid Sever | ity |
| Level and Treatment Arm | |
| Table 17: Summary of Primary Outcome (Relapse) by CTP | |
| Table 18: Summary of Relapse Status <sup>1</sup> for the Groups of Interest | |
| Table 19: Summary of Percent Days of Illicit Opioid Use <sup>1</sup> for Groups of Interest | 70 |
| Table 20: Summary of Abstinent Days <sup>1</sup> for Groups of Interest | 71 |
| Table 21: Summary of Number of Visits 'Present and Clean' for Groups of Interest | 72 |
| Table 22: Summary of Number Completing 24 Weeks of Treatment <sup>1</sup> for the Groups of Int | erest73 |
| Table 23: Summary of Trails A and B by Treatment Arm | 74 |
| Figure 10: Boxplots of Trails A by Treatment Arm | 75 |
| Figure 11: Boxplots of Trails B by Treatment Arm | 76 |
| Table 24: Summary of Stroop Color and Word Scores by Treatment Arm | 77 |
| Figure 12: Boxplots of Stroop Word Score by Treatment Arm | 78 |
| Figure 13: Boxplots of Stroop Color Score by Treatment Arm | 78 |
| Figure 14: Boxplots of Stroop Color-Word Score by Treatment Arm | 78 |
| Table 25: Summary of Subacute Withdrawal per HAM-D Items by Treatment Arm | 79 |
| Figure 15: Boxplots of HAM-D Score by Treatment Arm | 81 |
| Table 26: Summary of Subacute Withdrawal per SOWS Items by Treatment Arm | |
| Figure 16: Boxplots of SOWS Score by Treatment Arm | 84 |
| Table 27: Summary of Opioid Craving Items by Treatment Arm | 85 |
| Figure 17: Boxplots of VAS Score by Treatment Arm | |
| Table 28: Summary of Self-Reported Alcohol Use by Treatment Arm | |
| Table 29: Summary of Self-Reported Other Drug Use by Treatment Arm | |
| Table 30: Summary of Self-Reported Tobacco Use by Treatment Arm | |
| Table 31: Summary of Problems Related to Drug Abuse by Treatment Arm | |
| Table 32: Summary of HIV Risk by Treatment Arm | |
| Table 33: Summary of Treatment Emergent* Adverse Events by Treatment Arm | |
| rabio 55. Caminary of Froatmont Emorgonic Advolute Evento by Freatmont Alli | 100 |

| Table 34: Summary of Treatment Emergent* Serious Adverse Events by Treatment Arm110 |
|---|
| Table 35: Summary of Treatment Emergent* MedDRA Coded Adverse Events by Treatment |
| Arm111 |
| Table 36: Summary of Treatment Emergent* MedDRA Coded Serious Adverse Events by Treatment Arm117 |
| Table 37: Listing of Treatment Emergent* Adverse Events by Treatment Arm119 |
| Table 38: Listing of Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm120 |
| Table 39: Listing of Non-Treatment Emergent Adverse Events Among Screen Failures122 |
| SAE Narratives123 |
| Table 40: Listing of Serious Adverse Events by Treatment Arm124 |
| Table 41: Listing of Deaths by Treatment Arm125 |
| Table 42 Listing of Participants with HAM-D and/or CHRT Assessment Question Responses |
| Indicating Potential Suicidality by Treatment Arm126 |
| Table 43: Summary of Participants with Reponses Indicating Potential Suicidality by Treatment Arm128 |
| Figure 18: Participant-level Plot of HAM-D Question 3: Suicide by Treatment Arm 129 |
| Figure 19: Participant-level Plot of CHRT Question 14: I have been having thoughts of killing myself, by Treatment Arm |
| Figure 20: Participant-level Plot of CHRT Question 15: I have been having thoughts of how I might kill myself, by Treatment Arm |
| Figure 21: Participant-level Plot of CHRT Question 16: I have a plan to kill myself, by Treatment Arm |
| Figure 22: Participant-level Trajectories for Participants with Aspartate Aminotransferase > 225 IU/L by Treatment Arm |
| Figure 23: Participant-level Trajectories for Participants with Alanine Aminotransferase > 225 IU/L by Treatment Arm |
| Table 44: Listing of Liver Function Tests for ALT and AST exceeding 45 IU/L by Treatment Arm |
| Table 45: Summary of Injection Site Abnormalities by CTP |
| Table 46: Listing of Injection Site Abnormalities140 |
| Table 47: Summary of Withdrawal Symptoms (SOWS Composite Score) at Induction by |
| Treatment Arm |
| Table 48: Listing of Pregnancies by Treatment Arm |
| Live Birth Narratives |
| Table 49: Summary of Protocol Deviations in Randomized Participants, by Treatment Arm146 |
| Table 50: Summary of Protocol Deviations Among Screen Failures |
| Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category149 |
| Table 52: Listing of Protocol Deviations among Screen Failures by Deviation Category155 |

#### LIST OF ABBREVIATIONS

**Abbreviation Definition** AE Adverse Event

ALT Alanine Aminotransferase
ASI-Lite Addiction Severity-Index-Lite
AST Aspartate Aminotransferase

BMI Body Mass Index
BP Blood Pressure
BUP Buprenorphine

BUP-NX Buprenorphine+Naloxone (Suboxone®)
CAP College of American Pathologists
CCC Clinical Coordinating Center

CCC Clinical Coordinating Center
CFR Code of Federal Regulations
CHRT Concise Health Risk Tracking

CLIA Clinical Laboratory Improvement Amendment of 1988

CNS Central Nervous System
CoC Certificate of Confidentiality

CRF Case Report Form CTN Clinical Trials Network

CTP Community Treatment Program
DEA Drug Enforcement Agency

DHHS Department of Health and Human Services

DSC Data and Statistics Center

DSM-5 Diagnostic and Statistical Manual of Mental Disorders Fifth Edition

DSMB Data and Safety Monitoring Board
eCRF Electronic Case Report Form
EDC Electronic Data Capture
ERC Ethics Review Committee
FDA Food and Drug Administration

FTND Fagerström Test for Nicotine Dependence

FWA Federal Wide Assurance
GCP Good Clinical Practice
HAM-D Hamilton Depression Scale
HBsAB Hepatitis B surface antibody
HBsAG Hepatitis B surface antigen

HCV Hepatitis C Virus

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

HR Heart Rate

IND Investigational New Drug IRB Institutional Review Board

IM Intramuscular IV Intravenous

LFTs Liver Function Tests (AST, ALT, albumin and bilirubin)

LI Lead Investigator MD Medical Doctor

MDMA Methylenedioxymethamphetamine (Ecstasy)
MedDRA The Medical Dictionary for Regulatory Activities

Mg Milligrams

# **LIST OF ABBREVIATIONS (cont.)**

| Abbreviation | Definition |
|--------------|------------|
|--------------|------------|

MM Medical Management MOP Manual of Operations NDA New Drug Application

NIAAA National Institute on Alcohol Abuse and Alcoholism

NIDA National Institute on Drug Abuse NIH National Institutes of Health

NMS Non-Study Medical and Other Services

NP Nurse Practitioner

NTX Naltrexone NX Naloxone

OHRP Office for Human Research Protections

PA Physician Assistant
PI Principal Investigator
PLG Polylactide-co-glycolide
QA Quality Assurance

RAB Risk Assessment Battery

RAP-C Research Advisory Panel of California
RRTC Regional Research and Training Center

SAE Serious Adverse Event

SC Subcutaneous

SOWS Subjective Opiate Withdrawal Scale

TAU Treatment as Usual
TLFB Timeline Follow-Back
UDS Urine Drug Screen
VA Veterans Administration
VAS Visual Analog Scale

XR-NTX Extended-Release Naltrexone (Vivitrol®)

#### 1.0 INTRODUCTION

# 1.1 Study Objective

The primary goal of the study is to estimate the difference, if one exists, between XR-NTX and BUP-NX in the distribution of the time to relapse (i.e., loss of persistent abstinence) during the 6-month trial. Secondary objectives are to: (1) compare outcome on XR-NTX versus BUP-NX across a range of clinical safety and secondary efficacy domains, (2) explore demographic, clinical, and genetic predictors of successful treatment and moderators of differential effectiveness (i.e., what variables may help clinicians choose which of these treatments is best for a given patient), and (3) collect a limited dataset to permit analyses of economic costs and benefits of the two treatments.

# 1.2 Study Design

This is a multi-center, two-arm, 6-month (24-week), parallel-group, open-label, randomized controlled trial to examine the comparative effectiveness and safety of XR-NTX versus BUP-NX. Candidates will be individuals seeking treatment for opioid dependence (heroin or prescription opioids) who are admitted to an inpatient (detoxification and/or short term residential treatment) program for treatment of substance dependence. The study will be conducted in approximately 8 CTPs that: (a) provide opioid detoxification services (inpatient/residential), (b) have the capacity to maintain participants opioid-free, (c) have the capacity to initiate patients onto XR-NTX or BUP-NX. (d) have the capacity to maintain participants on XR-NTX or BUP-NX for the duration of the 24-week trial, (e) have a sufficient flow of patients completing detoxification and who do not routinely receive long-term medication-assisted therapy as to provide a sufficient population of potential participants to achieve study enrollment goals, and (f) can provide a minimum level of outpatient care (at least one group and/or individual counseling session per week) for 24 weeks. Candidates will be consented, screened, and randomized at the time of admission, during detoxification or during early abstinence. Participants meeting all eligibility criteria will be randomized to one of two treatment conditions, XR-NTX or BUP-NX. Treatment will be for 24 weeks in the context of a protocol-directed medical management treatment program and individual or group psychosocial counseling. Research visits will occur weekly for collection of urine samples and safety and other assessments. XR-NTX will be administered by injection on an approximately every-four-week basis; BUP-NX will be provided for take-home, initially on a weekly basis, transitioning to an every-two-week and then to an every-four-week schedule. Medical management for both conditions will be on a similar (weekly, transitioning to every-two-weeks, to every-four-weeks) schedule. The primary outcome measure will be the time to the event of relapse. XR-NTX will be provided as Vivitroi<sup>®</sup>. BUP-NX will be provided as Suboxone® film.

The Protocol will proceed in four phases.

Phase 1: Informed Consent, Screening, and Randomization (Days -15 through Day 0): This phase begins with informed consent during the index admission, and initiates enrollment, the conduct of all study-specific procedures and the collection of study data. During the first several days of an index admission, clinical and/or research staff will provide information about the study to potential participants (for scheduled admissions this information may be provided in advance of the admission). Guidelines for opioid detoxification are provided in the study MOP; data on detoxification utilization will be collected. This phase may take place from 1 day to 15 days. Following final review and confirmation of all eligibility criteria, randomization may proceed. Randomization may take place on the same day as informed consent and screening if recent liver function results are available, but in most cases will likely take place 2 or 3 days

later. Regardless of when randomization takes place, the date of randomization will be defined as "Day 0".

<u>Phase 2: Induction (Day 0 through Day 156)</u>: Following randomization, participants will be inducted onto their assigned active medication condition and treated as outpatients for 24 weeks per protocol. Guidelines for induction onto XR-NTX and onto BUP-NX are provided in the study MOP. Following induction, XR-NTX will be administered by injection approximately every 4 weeks; and BUP-NX will be quickly titrated upwards to maintenance doses. Induction should occur as soon as practicable following randomization, but may occur as late as week 22. Participants will continue into Phases 3 and 4 for research visits, even if not yet inducted onto their assigned medication.

Phase 3: Active Treatment (Week 1 through Week 24): Following randomization, participants will be inducted as soon as practicable and treated per their assigned active medication condition and followed as outpatients until 24 weeks post-randomization. Assessment visits will occur weekly. Participants whose induction onto their assigned study medication is delayed will also attend weekly research visits. Medical management visits will initially occur weekly, transition to every two weeks and then to every four weeks. In order to retain participants in treatment, and consistent with good practice, we permit flexibility with dosing. The window for Visit 1 is -3/+6 days to accommodate induction; however, induction may occur after Visit 1. A +/-3-day window will be permissible for subsequent weekly visits. For participants who relapse and/or become lost to follow up, a -3/+28 day window is permissible to complete the EOT visit. Participants who relapse will discontinue study medication and weekly research visits, but should be encouraged to attend the week 24 and follow up visits at weeks 28 and 36.

Phase 4: Post Treatment Follow-up (Week 25 through Week 36): Toward the end of the 24-week treatment period, participants will be referred for follow-up care in the community (which could include continuation of medication, if available, indicated, and desired), and follow-up outcomes will be assessed at week 28 and week 36 post-randomization. For participants receiving BUP-NX, who do not wish to continue, or for whom community resources are not available, the study will provide a two-week BUP-NX taper (beginning at the week 24 visit). A -3/+28 day window will be permissible for the scheduled week 28 visit and a +/- 4 week window will be permissible for the scheduled week 36 visit.

#### 1.3 Treatment Initiation

To maximize generalizability, this study has been designed to permit entry of participants throughout opioid detoxification and early abstinence. While XR-NTX can only be administered to individuals who have completed detoxification, the percentage of participants who are randomized early that are able to successfully initiate antagonist therapy is unknown. A risk to this study plan is that a differentially large percentage of individuals may be unable to initiate XR-NTX versus buprenorphine therapy.

#### 1.3.1 Study Data Analysis Modification

Timing of the randomization is important to execution of the design and may also be an important prognostic variable. All cases are classified into one of three groups at the time of randomization, those:

- (a) randomized within 24 hours of last (licit or illicit) opioid use;
- (b) randomized between 24 and 72 hours following last (licit or illicit) opioid use;
- (c) randomized more than 72 hours following last (licit or illicit) opioid use.

Each of these groups represents different clinical scenarios commonly encountered in CTN CTPs. Group (a) represents early decision-making, at such a time as to avoid unnecessary detoxification for those choosing BUP-NX. For group (b), decision-making occurs later during

detoxification, but while participants still need to surmount the detoxification hurdle to begin XR-NTX. Group (c) includes participants who can be readily inducted onto either medication.

Individuals in groups (a) and (b) comprise the early randomizers. A data analysis modification (assessment of whether the early vs. late randomizers have a differential treatment effect and if so, time to relapse will be estimated for early and late randomizers separately) will occur if differential treatment initiation is a problem for early randomizers (i.e., significantly fewer early randomizers are able to complete detoxification and XR-NTX induction. This assessment will occur after the entry of 100 cases randomized early in the detoxification process.

#### 1.4 Database Sources

Completed forms and electronic data will be entered into the data management system in accordance with the CRF Completion Guidelines established by the DSC. Only authorized individuals shall have access to electronic CRFs.

#### 1.5 Randomization

Immediately following the final assessment of eligibility, participants will be randomly assigned to one of the two conditions: XR-NTX or BUP-NX. Random assignment will be on a 1:1 ratio to one of the two conditions. A restricted randomization plan will be used with centralized, automated, randomized block assignments. Randomization will be stratified by two factors, site and pre-detoxification level of opioid use. While there will be important and otherwise uncharacterized differences between sites − including state and local treatment service environments, opioid misuse epidemiology, and patient-level customs regarding treatment, medications, and clinical trial participation − the level of heroin and other opioid use will likely be an important independent predictor of treatment retention and rates of negative urines as has been demonstrated in recent analysis of naltrexone opioid trials(Sullivan et al 2006; Carpenter et al 2009; Brooks et al 2010). The level of opioid use at treatment entry is a binary classification, operationally defined as 6 or more bags (or equivalent) IV heroin per day (<6 bags/day) or other routes of administration or other opioids.

Eligible participants will be randomized in a 1:1 ratio to the BUP-NX and XR-NTX arms. The randomization process will be performed by computer at a centralized location. Randomization will be stratified by site and pre-detoxification level of opioid use [6 or more bags (or equivalent) IV heroin per day (≥6 bags/day) over the 7 days prior to entry into the treatment program versus less than 6 bags (or equivalent) IV heroin per day (<6 bags/day) or other routes of administration or other opioids]. The block size chosen will be adequate to ensure approximate treatment balance. The number in each treatment group will never differ by more than a factor of KB/2 where B is the block size and K is the number of strata.

The randomization procedure will be conducted in a centralized process through the Clinical Trials Network (CTN) Data and Statistics Center (DSC). The DSC statistician will generate the randomization schedule using balanced blocks of varying sizes within strata to ensure lack of predictability along with relative equality of assignment across treatment groups. The DSC statistician will review randomization data on a regular basis to ensure that the scheme is being implemented according to plan. A randomization slot, once used, will not be re-allocated. Details of the randomization process are described in a separate Randomization Plan.

#### 1.6 Study Population

Study participants will be approximately 600 treatment-seeking heroin- and/or prescription opioid-dependent volunteers, without chronic pain requiring opioid therapy, who are willing to accept "agonist-based" or "antagonist-based" therapy. Randomization will be stratified by (1)

treatment site, and (2) baseline opioid use (high level use [≥6 bags {or equivalent} IV heroin/day] vs. all others [i.e., <6 bags {or equivalent} IV heroin/day and other routes of administration or other opioids]).

#### 1.6.1 Inclusion Criteria

- 1. Male or female;
- 2. 18 years of age and older;
- 3. Meet DSM-5 criteria for opioid-use disorder (heroin and/or prescription opioids);
- 4. Have used opioids other than as specifically prescribed within thirty days prior to consent:
- 5. Seeking treatment for opioid dependence and willing to accept "agonist-based" or "antagonist-based" therapy;
- 6. In good-enough general health, as determined by the study physician on the basis of medical history, review of systems, physical exam and laboratory assessments, to permit treatment with XR-NTX or BUP-NX;
- 7. Able to provide written informed consent;
- 8. Able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study;
- 9. If female of childbearing potential, be willing to practice an effective method of birth control for the duration of participation in the study.

#### 1.6.2 Exclusion Criteria

- 1. Serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make study participation hazardous to the participant or compromise study findings or would prevent the participant from completing the study. Examples include:
  - (a) Disabling or terminal medical illness (e.g., uncompensated heart failure, cirrhosis or end-stage liver disease) as assessed by medical history, review of systems, physical exam and/or laboratory assessments;
  - (b) Severe, untreated or inadequately treated mental disorder (e.g., active psychosis, uncontrolled manic-depressive illness) as assessed by history and/or clinical interview:
  - (c) Current severe alcohol, benzodiazepine, or other depressant or sedative hypnotic use likely to require a complicated medical detoxification (routine alcohol and sedative detoxifications may be included);
- 2. LFTs (ALT, AST) greater than 5 times upper limit of normal;
- 3. Suicidal or homicidal ideation that requires immediate attention;
- 4. Known allergy or sensitivity to buprenorphine, naloxone, naltrexone, polylactide-coglycolide, carboxymethylcellulose, or other components of the Vivitrol® diluent;
- 5. Maintenance on methadone at doses of 30mg or greater at the time of signing consent:
- 6. Presence of pain of sufficient severity as to require ongoing pain management with opioids;
- 7. Pending legal action or other reasons that might prevent an individual from completing the study;
- 8. If female, currently pregnant or breastfeeding, or planning on conception;

9. Body habitus that, in the judgment of the study physician, precludes safe intramuscular injection of XR-NTX (e.g., BMI>40, excess fat tissue over the buttocks, emaciation).

#### 2.0 OUTCOMES

# 2.1 Primary Outcome

The primary outcome measure will be the time to the event, with the event called relapse. By definition individuals are abstinent at the time of randomization. Relapse occurs if the participant is using any non-protocol prescribed opioids regularly starting at day 21 post-randomization or thereafter. Operationally, loss of persistent abstinence is defined as either: (a) four consecutive opioid use weeks, or (b) seven consecutive days of use by self-report. A use week is defined as any week during which a participant self-reports at least one day of use during that week, provides a urine sample positive for non-protocol opioids, or fails to provide a urine sample. Self-report of opioid (heroin or prescription opioids) and other substance use will be ascertained at each weekly study visit using the Time Line Follow-back for each day leading back to the previous visit. Urine will be collected at each study visit and tested for opioids. In the event that a participant reports no use, but their urine test indicates use, then we will regard the week as a use week. Missing urine samples will be classified as positive. The time of the event occurs at the start of the qualifying clinical event period (e.g., first of the 7 consecutive use days or start of the 4 consecutive weeks of use).

### 2.2 Secondary Outcomes

| Table 1: Protocol Secondary Outcomes and Hypotheses | |
|---|---|
| Outcomes | Hypotheses |
| Proportion successfully inducted onto assigned study medication (binary: did or did not receive first dose of XR-NTX, or achieve maintenance dose of BUP-NX) | BUP-NX will produce higher rate of successful induction than XR-NTX Significance/Rationale: XR-NTX induction requires completion of detoxification, whereas BUP-NX induction only requires onset of withdrawal symptoms. Thus XR-NTX may have more dropouts after randomization but prior to XR-NTX induction. |
| Adverse Events related to study medications | XR-NTX and BUP-NX will produce equivalent rates of SAEs, and equivalent rates of AEs, though AE pattern will differ somewhat (e.g. injection site reactions with XR-NTX) Significance/Rationale: Careful documentation of SAEs and AEs, including overdose episodes, would be considered essential safety data, and important component of a comparative effectiveness trial. |
| Opioid abstinence over time while on study medication (Weekly TLFB, confirmed by urine drug screens) | XR-NTX will produce greater opioid abstinence than BUP-NX Significance/Rationale: XR-NTX produces complete blockade of opioid effects, so that during treatment with monthly injections, opioid use can be expected to be minimal. In contrast BUP-NX may not produce complete blockade, or patients may reduce or stop doses for a few days and substitute other opioids (heroin, prescription opioids). |

| Table 1: Protocol Secondary Outcomes and Hypotheses | |
|---|---|
| Outcomes | Hypotheses |
| Alcohol and other drug use, over time (TLFB and UDS) | XR-NTX will be superior to BUP-NX in producing abstinence from alcohol and other drugs |
| | Significance/Rationale: Clinical trials show XR-NTX is effective for treatment of alcohol dependence, and naltrexone has some evidence of efficacy for stimulant dependence. |
| Cigarette smoking (FTND,<br>Tobacco Use Questionnaire,<br>VAS nicotine craving) | XR-NTX will reduce cigarette smoking compared to BUP-NX Significance/Rationale: Naltrexone has been studied as a treatment for nicotine dependence, with some support from clinical trials, although inconsistent. Given high morbidity and mortality associated with nicotine dependence, a comparative advantage of one or the other of these treatments at reducing smoking would be valuable to examine. |
| Opioid Craving (VAS) over time | XR-NTX will be superior to BUP-NX in reducing opioid craving Significance/Rationale: Krupitsky et al (Lancet 2011) pivotal XR-NTX trial showed, surprisingly, that XR-NTX reduced craving substantially compared to placebo. |
| Subacute withdrawal symptoms over time (HAM-D, SOWS) | XR-NTX will produce greater severity of subacute withdrawal symptoms than BUP-NX during the first month after randomization, but will be equivalent to BUP-NX in months 2 to 6 Significance/Rationale: Low-grade withdrawal-like symptoms (dubbed "naltrexone flu" by the Columbia group, and consisting typically of insomnia, fatigue, and anorexia, though not drug craving) have been observed in some patients in the 1 to 4 weeks after naltrexone initiation, resolving gradually. Further characterization of this syndrome would be important for developing treatment guidelines. |
| Problems related to drug abuse (ASI-Lite and EQ-5D) | XR-NTX will be superior to BUP-NX Significance/Rationale: Greater opioid and non-opioid abstinence on XR-NTX will result in fewer problems associated with active drug abuse. |

| Table 1: Protocol Secondary Outcomes and Hypotheses | |
|---|---|
| Outcomes | Hypotheses |
| HIV risk behavior over time (RAB and other HIV risk measures) | XR-NTX and BUP-NX will be equivalent Significance/Rationale: The opioid-dependent population is at high risk for HIV, both from injection drug use and from unsafe sexual practices. Effective treatment for the opioid dependence may reduce HIV risk behavior. Given the high morbidity and mortality associated with HIV, a comparative advantage of one or the other of these treatments would be valuable to examine. |
| Cognitive function (Trails<br>Making Test Parts A and B,<br>Stroop) | XR-NTX and BUP-NX will be equivalent Significance/Rationale: Some providers and policy-makers are concerned that patients maintained on BUP-NX will have opioid-agonist-related cognitive impairment. |

#### 3.0 GENERAL CONSIDERATIONS

#### 3.1 Terminations

There are multiple types of terminations in this study, end of study medication, medical management termination and study termination. Study medication will be discontinued in the event of intolerable side effects, safety concerns preventing further medication treatment (i.e., pregnancy), relapse, or the end of the 24-week active treatment phase. Participants discontinuing medication, but not yet meeting relapse criteria, prior to week 24 will continue within the same study assessment schedule. Participants meeting relapse criteria will discontinue medication, research visits and complete a medical management termination form. All participants who end treatment early (prior to week 21) will be encouraged to attend a visit at week 24 and will be seen in long-term follow-up (weeks 28 and 36). In all cases of treatment discontinuation, the research team will make an effort to arrange for continued community treatment, as appropriate and available, including further XR-NTX and BUP-NX, or methadone maintenance and intensive outpatient psychosocial aftercare. For participants receiving BUP-NX, who do not wish to continue, or for whom community resources are not available, the study will provide a two-week BUP-NX taper, if clinically appropriate.

Dropout from treatment is a typical failure mode for the treatment of opioid dependence with both XR-NTX and BUP-NX. A sensitivity analysis will be performed to examine the impact on the hazard ratio and its confidence limits of alternative endpoint definitions. In particular for the primary endpoint, individuals who withdraw will be considered events if they fail to provide weekly urine specimens. An alternative to the protocol definition which introduces these as censored observations will be examined. The analyses of these events can be complex as standard assumptions (missing at random) may not be plausible.

Other outcome variables (opioid and other substance use over time, craving, mood, etc.) will have missing data due to missed visits and dropout from treatment and from study participation. The generalized linear model, or mixed effects model frameworks that will be used for analyses, works with what data are gathered, and assumes missing data are missing at random. For selected secondary outcome analyses, sensitivity analyses will be considered to examine the stability of estimated treatment effects in the face of departures from the assumption of missing at random.

Aggressive tracking procedures will be put into effect to attempt to locate participants and reengage them, and to minimize missing data. These procedures will be detailed in the study MOP. The greatest likelihood of violation of the assumption of missing at random derives from dropouts, since participants assigned to XR-NTX may dropout from the study for different reasons than participants assigned to BUP-NX, creating the potential for differential attrition. Differential study attrition for the two treatment groups, where outcome differs between the dropouts is a threat to the validity of the outcome analysis. Minimizing the rate of study dropout and loss to follow-up, through aggressive tracking and follow-up, serves to reduce this threat. At a minimum the data gathered on dropouts can be used to test the assumption of missing at random, by examining whether dropouts from the different treatment assignments have similar or different outcomes.

# 3.2 Study Modification for Differential Treatment Initiation

To maximize generalizability, this study has been designed to permit entry of participants throughout the opiate detoxification process and early abstinence. At the time the study was designed, it was understood that community-based practice of detoxification and medication induction would vary across sites and across patients within sites. It was further decided that the

protocol would allow this variation in community based practice of detoxification-induction, consistent with the aims of an effectiveness trial to test the medications under real world conditions. It was also anticipated that induction onto BUP-NX would be easier than induction onto XR-NTX for patients who are randomized "early" while opioids are still in their system. This is because BUP-NX can be safely initiated while opioids are still in the system, as long as some signs of withdrawal begin to develop, while for XR-NTX one needs to wait until detoxification is completed. This delay is an opportunity for differential attrition between the 2 study arms. The concern is that a higher induction failure rate on XR-NTX, among those randomized early, will contribute to differences in outcome (time-to-relapse) across the 6 month trial, with induction failure leading to relapse. If this is the case, then the interaction between early vs. late randomization and treatment assignment on the primary outcome (time to relapse) becomes germane.

Therefore, after the entry of 100 "early randomizers" (as defined in Protocol Section 8.3 [or Section 1.5 above]) we will compare the induction success rate in these early randomizers on XR-NTX vs. BUP-NX with a test of difference between proportions. The decision rule has >80% power (alpha=2.5% 1 tail) to identify differences of .25 or greater if the true initiation rate for the BUP-NX is in the expected range (>=.85). If the difference in induction failure rate is statistically significant, then the following plan will be followed:

- 1. Increase the sample size to end enrollment at such time as 350 late randomizers have been enrolled to increase power to estimate the difference in primary outcome (time-to-relapse) in this late randomizer group. It is projected that at such time the total N will be approximately 600.
- 2. Amend the data analysis plan to incorporate an interaction term in the analysis model.

# 3.3 Sample Size and Power Calculations

The therapeutic strategies defined above will be evaluated and compared in a two-arm randomized open-label multi-center trial.

Original Projected Sample Size: 200 per treatment group. N = 400 total.

<u>Data Analysis Modification Projected Total Sample Size</u>: N~600 total sufficient to enroll 350 late randomizers.

Rationale: The primary outcome is the time to relapse as defined above. Meta-analyses of randomized controlled trials of BUP-NX maintenance treatment for opioid dependence suggest that approximately 50% of patients are retained in BUP-NX treatment with good clinical outcome over 6 months. (Mattick and Kimber 2008). Extended release naltrexone preparations have had few prior randomized comparisons but observations from a recent Russia-based trial evaluating the XR-NTX dose and formulation proposed for this trial had good results with 53% receiving all monthly injections and retained for 6 months. Direct randomized comparison of these approaches has not been performed.

We evaluate the anticipated variability of the primary terminal results by simulating under exponential distributional assumptions with event (relapse) grouping after the first 21 days and using proportional hazards without censoring. Let one treatment have a 6-month success rate of 40% with exponential failure. We use a lower success target than indicated in the above paragraph because the use of the early randomization time point is expected to increase the percentage of participants who are failures. There would be minimal impact on detectable alternatives if a higher 50% success rate was used. From the plot below, we observe that the 95% CI width for the hazard ratio for the 50<sup>th</sup> percentile of the simulation results under both the null and alternative hypotheses decreases by 31%, 19%, and 14% as the sample size increase

by 50/arm from a base of 50/arm. CI width decreases by 11% when the sample size increases from 200/arm to 250/arm. We have selected 200/arm as subsequent precision improvements with these criteria are close to 10% per 100 sampling units.

Beyond a sample size of 150 to 200 patients per group, further increments in sample size (200 per group, 250 per group, 300 per group, etc.) yield diminishing returns in terms of only relatively small further narrowing of the 95% confidence interval. The rationale for increasing the total sample size to N  $\sim$ 600, in the event of a significant difference in induction success rate among early randomizers, is that given the current ratio of early to late randomizers, N  $\sim$ 600 total will yield approximately 250 early randomizers and 350 later randomizers. 350 late randomizers (N = 175 per treatment group) is close to the 400 (N = 200 per group) originally planned, and will yield a very similar (only slightly wider) 95% confidence interval. This will preserve the intent to achieve a relatively precise estimate of the difference in relapse rates among late randomizers.

Figure 1: Simulation results for the 50th and Upper 95th percentile of the 95% Confidence Interval Widths for the Hazard Ratio, selected sample sizes with lambda=0 and lambda=0.678



The decision theoretic properties of n=200/arm is evaluated further under a decision theoretic approach and using the logrank test. With two-sided alpha = 0.05, N = 400 total participants provides 90% power to detect a hazard ratio of .63 for the second treatment. Table 2 provides additional characterization of power characteristics of the sample size.

| Table 2: Detectable Alternatives and Power for 2-tailed 5% level logrank test without censoring Null distribution has a 40% 6 month success rate, N1=N2=200 | |
|---|---|
| Power (%) Hazard Ratio 6 Month Survival Rate (%) under the Alternative | |
| 90.0 | .633 56.0 |
| 80.0 | .678 53.8 |

Note that inclusion of the baseline level of opioid dependence severity stratification variable in the statistical model as a covariate may increase power and narrow the confidence limits on treatment hazard ratios, should divergent success rates be present in the strata groupings.

Secondary analyses of moderators of treatment effect are important to trial sample size selection. With approximately 200 XR-NTX cases evenly split between two levels of a classifying variable, we would have 79% power to detect, using a two-tailed 5% level test of a binary endpoint, a 20 percentage point difference between the groups. Thus the selected sample size would be relatively robust in its ability to determine whether there are important differences in therapeutic success rates for major demographic or baseline clinical factors.

#### 3.4 Interim Analysis

The study will undergo safety monitoring by the designated DSMB. Both therapies are standard therapies with regulatory approval for treatment of opiate abuse. The treatment strategies have not been directly compared before and classic interim efficacy monitoring is not planned as both are considered acceptable therapies. An adaptive strategy for addressing substantial differential treatment initiation is described above and in Section 5.2.

#### 3.5 Software

All analyses will be performed utilizing SAS® version 9.3. All statistical tests will be conducted at the 5% Type I error rate (two-sided). When multiple tests are conducted, the chance of finding a significant difference in one of the tests, when in fact no difference exists, is greater than the stated Type I error rate. The investigators are aware of the multiple testing issues and will interpret results with caution and use confidence intervals where possible.

#### 3.6 Analysis Populations

Each primary and secondary efficacy outcome measure will be analyzed for the intent-to-treat (ITT) and evaluable population. The intent-to-treat principle is that participants will be analyzed in the groups to which they were randomized, regardless of whether they received the randomized study medication. Another analysis population of interest is the as-treated population. The as-treated population will consist of only participants who were inducted onto study medication.

Major differences in the results for the ITT and as-treated populations, if any, will be further explored. While there is every intention to be complete in describing the analyses to be performed, it is not possible to anticipate every contingency, and some adjustments may be required to meet constraints posed by the structure of the data. Constraints such as non-linearity, non-normality, etc. may lead to different but more appropriate approaches to analysis.

#### 3.7 Distributional Assumption Tests

Empirical distributions of all variables will be visually inspected to detect outliers. The underlying proposed statistical methods for each analysis will be examined, primarily through inspection of graphical displays, standardized residuals, or influence diagnostics. Where appropriate,

transformations will be utilized or analyses will be performed utilizing a more appropriate distribution.

# 4.0 ANALYSES OF DEMOGRAPHIC AND BASELINE DATA

CTN-0051: X:BOT

Statistical Analysis Plan

The demographic variables for this study include: gender, age, race, ethnicity, education level, employment status, and marital status. The baseline clinical characteristics include: opioid dependence severity, severity of other substance use, severity of mood/anxiety symptoms, severity of opioid withdrawal symptoms, current/past co-occurring psychiatric disorders, current medical disorders, select genetic markers, history of legal problems, currently under legal supervision (parole, probation or mandated).

Descriptive statistics for baseline and demographic variables will be presented for participants randomized to each of the treatment arms and overall. Descriptive statistics will include N, mean, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum for continuous variables and proportions and percentages for categorical variables. Since randomization is expected to produce balance at baseline between the two arms of the trial, statistical comparisons of treatment groups with respect to baseline characteristics will not be conducted. The updated CONSORT statement no longer recommends formal testing of statistical significance of differences between baseline characteristics.

#### 5.0 STATISTICAL ANALYSES

# **5.1** Timing of Randomization Definitions

The early randomizers are those participants randomized within 72 hours following the last licit or illicit opioid use. The late randomizers are those participants randomized greater than 72 hours following the last licit or illicit opioid use. To determine the timing of randomization, it is necessary to know the day and time (measured using 24 hour clock) of last licit or illicit opioid use. On rare occasions, missing values for one or both of these measures may exist. For primary analysis purposes, if the date of last licit or illicit opioid use is available but the time is not, the participant's time will be imputed to be 00:00. This will impute the longest potential time from randomization. If the date of last licit or illicit use is missing, the participant categorization will be imputed by the predominant proportion of the randomization timing status in that site.

# 5.2 Differential Treatment Initiation for Early Randomizers Assessment

The study modification assessment will be completed when the 100 participants who have been randomized within 72 hours following his/her last (licit or illicit) opioid use have had at least 21 days post-randomization to be inducted onto study medication. The analysis population for the early randomizers assessment will only consist of the first 100 early randomizers. The timing of the database freeze will ensure that these 100 early randomizers have had at least 21 days post-randomization to be inducted onto study medication.

#### 5.2.1 Induction Status Determination

A participant's induction status will be a binary variable of Yes or No. For the participants randomized to BUP-NX, participants will be defined as inducted onto the study medication if he/she has been dispensed medication as measured on the BUP-NX dose log; otherwise, the participant will be defined as not being inducted onto study medication. In a similar manner, for participants randomized to XR-NTX, participants will be defined as inducted onto the study medication if he/she has received an injection of the study medication. Note, the definition of induction status is not dependent upon the number of days for induction to occur.

#### 5.2.2 Induction Status Analysis

The null hypothesis is:

$$H_0: p_{XR-NTX} = p_{BUP-NX}$$
  
 $H_A: p_{XR-NTX} \neq p_{BUP-NX}$ 

Where  $p_{XR-NTX}$  is the proportion of early randomizer participants in the XR-NTX group who were

inducted and  $p_{BUP-NX}$  is the proportion of early randomizers participants in the BUP-NX group who were inducted. The Fisher's exact test will be used to determine statistical significance at a significance level of 0.05.

#### 5.3 Primary Outcome

The primary outcome measure will be the time to the event, with the event called relapse. By definition individuals are abstinent at the time of randomization. Relapse occurs if the participant is using any non-protocol prescribed opioids regularly starting at day 21 post-randomization or thereafter. Operationally, loss of persistent abstinence is defined as either: (a) four consecutive opioid use weeks, or (b) seven consecutive days of use by self-report. A use week is defined as any week during which a participant self-reports at least one day of use during that week, provides a urine sample positive for non-protocol opioids, or fails to provide a urine sample.

Self-report of opioid (heroin or prescription opioids) and other substance use will be ascertained at each weekly study visit using the Time Line Follow-back for each day leading back to the previous visit. Urine will be collected at each study visit and tested for opioids. In the event that a participant reports no use, but their urine test indicates use, then we will regard the week as a use week. Missing urine samples will be classified as positive. The time of the event occurs at the start of the qualifying clinical event period (e.g., first of the 7 consecutive use days or start of the 4 consecutive weeks of use).

# 5.3.1 Primary Outcome Criteria

Relapse assessment starts Day 21 post-randomization with the day of randomization as Day 0 and ends at the Week 24 visit. As noted above, relapse is defined in two ways:

#### a) Four consecutive opioid use weeks

- i) There are three ways that a use week can be established:
  - (1) Participant self-reports at least one day of use during that week

The self-report of use is measured between the weekly visits and thus does not always include the review of exactly seven days. At the weekly visit, if the previous visit was missed, the participant's daily self-report opioid use is assessed from the start of the current visit window (i.e. the beginning of the window as specified by the protocol calendar, see table below) to the day before the current visit. Conversely, if the previous visit was attended, the participants daily self-report opioid use is assessed from the previous visit attended day to the day before that current visit. Note, only participants self-report collected on or after Day 21 is used in evaluating whether the week is a use week. Thus, if the Week 3 visit is attended on Day 21, there cannot be a use week based on self-reported opioid use.

| Table 3: CTN-0051 Protocol Calendar | | | |
|---|---|---|---|
| Visit<br>Number | Target<br>Day | Beginning<br>Window<br>(Days) | End of<br>Window<br>(Days) |
| 00R | 00 | 00 | 00 |
| 01 | 06 | 3 | 12 |
| 02 | 13 | 10 | 16 |
| 03 | 20 | 17 | 23 |
| 04 | 27 | 24 | 30 |
| 05 | 34 | 31 | 37 |
| 06 | 41 | 38 | 44 |
| 07 | 48 | 45 | 51 |
| 08 | 55 | 52 | 58 |
| 09 | 62 | 59 | 65 |
| 10 | 69 | 66 | 72 |
| 11 | 76 | 73 | 79 |
| 12 | 83 | 80 | 86 |
| 13 | 90 | 87 | 93 |
| 14 | 97 | 94 | 100 |
| 15 | 104 | 101 | 107 |

| Table 3: CTN-0051 Protocol Calendar | | | |
|---|---|---|---|
| Visit<br>Number | Target<br>Day | Beginning<br>Window<br>(Days) | End of<br>Window<br>(Days) |
| 16 | 111 | 108 | 114 |
| 17 | 118 | 115 | 121 |
| 18 | 125 | 122 | 128 |
| 19 | 132 | 129 | 135 |
| 20 | 139 | 136 | 142 |
| 21 | 146 | 143 | 149 |
| 22 | 153 | 150 | 156 |
| 23 | 160 | 157 | 163 |
| 24 | 167 | 164 | 195 |

# (2) Participant provides a urine sample positive for non-protocol opioids

The urine drug screen (UDS) is used to assess whether the urine sample is positive for non-protocol opioids. Only UDSs assessed at weekly visits will be used to determine relapse status. UDSs assessed at the inductions that occur prior to Day 21, supplemental induction or end of treatment visits will not be used to assess relapse. Note, any induction UDSs that occur after Day 21 are entered into the weekly visit, and the results are duplicated in the induction visit UDS. Additionally, supplemental UDSs are not expected and should not be entered except for supplemental induction visits. If an out of window visit occurs, the UDS collected at that out of window visit will contribute to the use week calculation of that visit.

For the BUP-NX arm, use for a urine sample is defined as a positive result for any of the following tests: Opiates (2000 ng), Oxycodone (OXY), Methadone (MTD), or Opiates (300 ng). For the XR-NTX arm, use for a urine sample is defined as a positive result for any of the following tests: Opiates (2000 ng), Oxycodone (OXY), Methadone (MTD), Opiates (300 ng) or Buprenorphine (BUP).

# (3) Participant fails to provide a urine sample.

UDSs that are not collected, determined to be adulterated or out of the temperature range result in a use week. If the field indicating adulterated or out of temperature range is missing, that UDS would result in a use week. Additionally, missed visits are tracked using the missed visit form. If the missed visit form is completed, that week is designated a use week.

#### b) Seven consecutive days of use by self-report

The timeline follow back dataset is used to calculate the number of consecutive use days. A use day is defined as values for the opioids mentioned above. The first instance of seven consecutive days of use by self-report will define the participant as relapsed. The first day of the seven consecutive days is defined as the relapse start date.

#### 5.3.2 Determination of the Start of the Clinical Qualifying Event

For the purposes of the primary outcome analyses, the relapse start day will be used. The time of the event occurs at the start of the qualifying clinical event period (e.g., first of the 7 consecutive use days or start of the 4 consecutive weeks of use). If both of the criteria above (a and b) are met, then the earlier of the two relapse start dates will define the day that the relapse criterion met for the purposes of primary outcome analyses.

When a participant's data indicates four consecutive weeks of use, the reason the first week was defined as a use week will be used to determine the start of the qualifying clinical event period. The first use week could be due to either a self-report of at least one day of use, a urine sample positive for non-protocol opioids, failure to provide a urine sample or some combination of these reasons. The following table outlines how the start of the clinical qualifying event will be determined in the case of a participant having four consecutive weeks of use.

| Table 4: Determination of the Start of the Clinical Qualifying Event | | | |
|---|---|---|---|
| Reason for First Use Week | | t Use Week | |
| Missing<br>UDS | Positive<br>UDS | Self-report of<br>at least one<br>day | Start of the Clinical Event |
| * | | * | Date of first self-reported use |
| | * | * | Day of first self-reported use |
| | | * | Day of first self-reported use |
| | * | | Day of positive urine drug screen |
| * | | | First study day of the first use week period as defined by the protocol calendar |

#### 5.3.3 Primary Outcome Analysis Methods

Since the results of the interim analysis indicated a differential treatment initiation rate assessment, the data analysis modification will be employed. As noted in Section 3.2, if there is a differential treatment initiation rate in the early randomizers group, an interaction term for the treatment by randomization timing variables will be incorporated into the final analysis model.

Data will be analyzed using a Cox proportional hazards model. The model is as follows:

$$\log h(t \mid CUF) = \log h_0(t \mid CUF) + \beta_1 * Treatment + \beta_2 * TIMING + \beta_3 * CTP + \beta_4 * STRATA + \beta_5 * Treatment * TIMING$$

where h is the hazard rate, roughly defined as the probability per time unit that a case that has not relapsed to the beginning of the respective interval will relapse in that interval. Conceptually, it can be thought of as the number of relapse per time units in the respective interval, divided by the average number of non-relapse cases at the mid-point of the interval. The quantity h0 is an arbitrary baseline hazard rate.

The SAS PHREG procedure will perform survival analysis based on the Cox model to estimate the hazard ratio for the treatments. The 95% Wald Confidence limits will be estimated.

The following SAS Code will be used to analyze the data:

```
PROC PHREG;
CLASS TREATMENT (REF='BUP-NX') TIMING (REF='Late');
MODEL TIME*STATUS = TREATMENT TIMING CTP STRATA
TREATMENT*TIMING;
HAZARDRATIO TREATMENT;
RUN;
```

The variables included in the SAS code are described as follows:

- TREATMENT- This variable defines the randomized treatment assignment. (BUP-NX or XR-NTX)
- TIME- Time to relapse
- STATUS- Censoring variable
- CTP- CTP
- STRATA- Randomization Stratification factor pertaining to the baseline opioid severity level classified as <6 bags (Low Severity) or ≥ 6 bags (High Severity).
- TIMING- Binary baseline variable (early vs. later randomization as noted in Section 5.1 defined as either 'Late' or 'Early').

The initial analysis will be the construction of the asymptotic 95% CI for the hazard ratio of the difference between the treatment arms in the time to event distribution for the primary outcome. The study arm success rates with confidence intervals at week 24 and the difference in success rate at that time point and associated confidence intervals will be constructed.

If the data analysis modification is implemented, the binary baseline variable (early vs. later randomization as previously defined) is included in the primary outcome analysis (outcome = time-to-relapse) as a covariate, a priori. The early vs. late randomization covariate by treatment interaction is included in the primary outcome analysis. If the covariate (early vs. late randomization) by treatment interaction is significant at P < .10, then the interaction term is retained in the final model. To characterize the interaction, the effect of treatment assignment (which includes the interaction and the main effect for treatment) (i.e., the difference in time-to-relapse between treatments) is estimated separately in early vs. late randomizers, and these two separate estimates become the primary findings of the study. If the covariate (early vs. late randomization) by treatment interaction is not significant (p>=.10) then the interaction term will be removed from the model and the main effect estimate will be the primary finding of the study. Exploratory analyses will also evaluate whether the primary outcome measure of time-to-relapse is associated with the number of hours between last licit or illicit opioid use and randomization, that is, a continuous measure of the randomization timing. Both linear and non-linear effects will be explored as potential effect modifiers.

The Cox proportional hazard model is based on the following assumptions. First, there is a proportional hazards assumption, such that if an individual has a risk to opioid use at initial time point that is twice as high as that of another individual, then at all later times the risk of opioid use remains twice as high. Secondly, factors such as the way participants are recruited into a study and the determination of relapse remains constant over the period of the study i.e. censoring should be independent of an event (relapse) happening. The proportional hazards assumption will be assessed by testing of the time to relapse variable and the corresponding covariates of interest. If the proportional hazards assumption is not met, the final model will incorporate a time-dependent variable for the non-proportional predictors in the Cox model.

# 5.4 Secondary Analyses of Primary Outcome Measure

Subsequent analyses will explore the treatment effect as a function of time, stratification variables and other factors that may have differential impact on treatment success. The analyses will first model the time to event primary outcome measure as a function of treatment assignment (XR-NTX vs. BUP-NX), opioid dependence severity stratum, site, and the two way treatment interaction terms (site by treatment and stratum by treatment) in a proportional hazards regression model. The Cox model previously described in the primary outcome analysis can separately incorporate covariates that are fixed (at baseline). The constancy of the relative hazard assumption will be examined via the interaction of treatment and time, and the interaction between treatment and baseline severity will be tested.

If treatment by site interaction is significant, we will further investigate if the interaction is quantitative or qualitative. A quantitative interaction between treatment and site will indicate that the treatment differences are in the same direction across sites but the magnitude differs from site to site, while a qualitative interaction reveals that substantial treatment differences occur in different directions in different sites. As indicated by Gail and Simon (1985), the existence of a quantitative interaction between treatment and site does not invalidate the analysis in pooling data across centers. Hence we will analyze the data ignoring the treatment-by-site interaction. But when there is a qualitative interaction the treatment effect itself would not make any sense and any kind of analysis claiming a common treatment effect will be questionable.

If the stratum by treatment interaction has a p-value <0.10, then this will be taken to indicate differences in strata-specific efficacy. We note that if this interaction is qualitative (i.e., reversal of treatment advantage in the subgroups) this will have important consequences for future treatment and research decisions. We will test the pair-wise differences between XR-NTX and BUP-NX, separately in the low dependence vs. high dependence subgroups, and further examine the differences with an ordinal/continuous dependence covariate. Note that we are not powering the study to detect the interaction; however, given the likelihood that baseline use predicts outcome, or may interact with treatment (Nunes et al 2011), the coefficient of the main effect of treatment in the model is not meaningful in the presence of an interaction with baseline covariates, and that a significant interaction should prompt testing of the region(s) of the baseline covariate where the probability of treatment successes differ (Nunes et al 2011; Pocock et al 2002).

Secondary analyses of the 24 week successes will include screening baseline variables to identify potential subgroups in the treatment groups with differential results.

All participants who were randomized will be included in the primary efficacy analysis. Note that the primary analysis for the time to relapse inference is based on the assumption that all missing UDSs' are positive.

A secondary analysis of the primary outcome measure will also be presented assuming these observations are censored which will allow us to assess robustness of conclusions to the deviation from the MAR missing data assumption. See Section 6.0 for additional details.

Summary statistics for the primary outcome measure will be provided for each CTP.

### 5.5 Secondary Outcomes

Most secondary outcome analyses will follow a similar form and strategy to that above, with different linear models as appropriate for the form of the secondary outcome variable: dichotomous secondary outcomes will use logistic regression; time-to-event variables will use survival analysis with Cox models; continuous variables or count variables (e.g., bags per day of heroin use) will use mixed effect models depending on the distribution of the outcome (e.g., normal, Poisson, negative binomial, zero-inflated). Repeated measures will have time in the model in addition to treatment and baseline covariates.

For the secondary outcome measures that are continuous a mixed effects model will be used to analyze the data incorporating appropriate covariates. The model for secondary outcomes that are continuous can be explained in matrix form as follows:

$$\mathbf{y} = \mathbf{X}\boldsymbol{\beta} + \mathbf{Z}\mathbf{b} + \varepsilon$$
$$\mathbf{b} \sim N_q(0, \Psi)$$
$$\varepsilon \sim N(0, \sigma^2 I)$$

Where

- y is the N (sample size) × 1 secondary outcome vector.
- **X** is the N × p model matrix for the fixed effects (e.g. Treatment).
- $\beta$  is the p × 1 vector of fixed-effect coefficients.
- **Z** is the N × q model matrix for the random effects (e.g. Site).
- **b** is the q × 1 vector of random-effect coefficients.
- $\varepsilon$  is the N × 1 vector of errors for outcome.
- $\psi$  is the g × g covariance matrix for the random effects.
- $\sigma^2 I$  is the N × N covariance matrix for the errors.

#### 5.5.1 Induction Success

Successful initiation of protocol medication is an important binary outcome that may also be useful to subsequently explain differences in the primary outcome. The induction success outcome will be defined as noted in Section 5.3.1. Data will be analyzed using a logistic regression model. The model will include variables for treatment arm, a continuous measure of the randomization timing and the corresponding interaction term. The continuous measure of randomization timing will be the number of days between randomization and last licit or illicit use of opioids.

#### 5.5.2 Opioid Abstinence

Opioid abstinence will be measured using the TLFB and confirmed by urine drug screens.

#### 5.5.3 Cigarette Smoking

Cigarette smoking is assessed by the FTND, Tobacco Use Questionnaire and visual analog scale for nicotine craving assessments.

The visual analog scale for nicotine craving is assessed at multiple follow-up timepoints and thus a mixed effects model will be used to assess whether there is a treatment effect with respect to the VAS nicotine craving scale.

#### 5.5.4 Opioid Craving

Participants' cravings for opioid craving is documented on visual analog scales (VAS) via scores that range from 0 (no craving) to 100 (most intense craving possible). The VAS assessing opioid craving is completed at each study visit throughout the active treatment phase. A mixed effects model analysis will be conducted with treatment as a covariate.

#### 5.5.5 Subacute Withdrawal Symptoms

Subacute withdrawal symptoms are measured by the HAM-D and the SOWS.

# 5.5.6 Drug Use Problems

There are two assessments that capture data on drug use problems, the ASI-Lite and the EQ-5D.

The ASI-Lite is derived from the Fifth Edition of the ASI, a structured clinical interview that yields scores for seven areas of functioning typically impacted by addiction, including medical status, employment status, drug use, alcohol use, family status, legal status, and psychiatric status. Opioid use questions, including the main type of opioid used by the participant, whether a prescription opioid or heroin, the onset of the use, the participant's perception of the substance that is most problematic, and their present treatment goal will also be assessed at screening as part of the ASI assessment. The ASI-Lite is completed at baseline, at the end-of-treatment visit (week 24/EOT), and at the week 36/EOS follow-up visit.

The seven areas of functioning measured by the ASI-Lite will be analyzed using a mixed effects model with treatment as a covariate. These seven tests will be performed without adjustment for multiple testing.

# 5.5.7 HIV Risk Behavior as Assessed by the RAB

The sex risk scale of the RAB, which produces a score ranging from 0-28, will be considered as a continuous response variable, and treatment effect will be analyzed using mixed effects model.

#### 5.5.8 Cognitive Function

The Trails Making test Parts A and B and the Stroop test will be used to assess cognitive function.

# 5.6 Minority/Gender Analyses

In accordance with NIH guidelines, repeated Cox regression model analyses will be completed to determine whether treatment response was significantly affected by participant minority/gender status using an interaction term for treatment and minority/gender as appropriate.

#### 6.0 MISSING DATA

The primary outcome in this study defines missing urines as positive opioid use. Thus, missing value imputation of the urine drug screens is not necessary for the purposes of the primary outcome.

Dropout from treatment is a typical failure mode for the treatment of opioid dependence with both XR-NTX and BUP-NX. A sensitivity analysis for the primary outcome analysis will be performed to examine the impact on the hazard ratio and its confidence limits of alternative endpoint definitions. In particular for the primary endpoint, individuals who withdraw will be considered events if they fail to provide weekly urine specimens. An alternative to the protocol definition which introduces these as censored observations will be examined. The analyses of these events can be complex as standard assumptions (missing at random) may not be plausible.

Other outcome variables (opioid and other substance use over time, craving, mood, etc.) will have missing data due to missed visits and dropout from treatment and from study participation. The generalized linear model, or mixed effects model frameworks that will be used for analyses, works with what data are gathered, and assumes missing data are missing at random. For selected secondary outcome analyses, sensitivity analyses will be considered to examine the stability of estimated treatment effects in the face of departures from the assumption of missing at random.

#### 7.0 SAFETY ANALYSES

#### 7.1 Physical Examination

The study clinician will complete a physical examination, including blood pressure and heart rate, to ensure that there are no medical concerns regarding participation and to gather baseline information regarding the participant's physical health. During the screening physical exam, a description of the participant's body habitus will be documented and the study clinician will examine the planned injection sites to ensure adequacy for XR-NTX gluteal intramuscular injection of naltrexone with the supplied needle. The physical examination will be performed at screening and will be repeated at the end-of-medication visit (if medication is stopped early) or at the end-of-treatment visit (week 24). The physical exam, blood pressure and/or heart rate may be repeated at MM visits at the discretion of the medical clinician.

# 7.2 Concise Health Risk Tracking-Self Report (CHRT-SR)

The CHRT-SR (Trivedi 2011) is a 16-item participant self-report assessment of suicidality and related thoughts and behaviors. The scale is designed to quickly and easily track suicidality in a manner consistent with the Columbia Classification Algorithm of Suicide Assessment (C-CASA) S(Posner 2007). The CHRT-SR will be assessed at screening, induction, at subsequent MM visits and at the week 28 and 36/EOS visits. The CHRT-SR will assess high risk suicide ideation by a positive response (Agree or Strongly Agree) on any of the last three questions (thoughts of, thoughts of how and/or a specific plan to commit suicide) and prompt a clinician assessment for suicide risk before leaving the clinic.

#### 7.3 The Hamilton Depression Scale (17 item) (HAM-D)

The 17-item Hamilton Depression Scale (HAM-D) is a clinician-administered instrument, useful for following both depression and suicidal ideation, and also for following typical symptoms of subacute withdrawal (e.g., low appetite, fatigue, poor sleep). For the purpose of this study, adequately trained research staff conduct the Hamilton Depression Scale (HAM-D).

The HAM-D is completed at screening, at weeks 1, 2, 3, 4, 8, 12, 16 and 20, at the end-of-treatment visit (week 24/EOT), and at each follow-up. A score of 1 or more to item 3 (suicidality) prompts a clinician assessment for suicide risk before leaving the clinic. Summaries of the suicidality question are tabulated for the purposes of safety analyses.

The HAM-D score is calculated by summing the first 17 items on the HAM-D form. A sum of 0 to 7 is considered to be normal, 8 to 13 is defined as mild depression, 14 to 18 as moderate depression, 19 to 22 as severe depression, and greater than or equal to 23 is defined as very severe depression.

# 7.4 Clinical Laboratory Tests

Liver function tests (LFTs, consisting of AST, ALT, albumin and bilirubin) and urine pregnancy test (for females) will be performed to help determine eligibility at screening. Receipt and review of laboratory test results is necessary before confirming eligibility, conducting randomization and starting study medication. Results of LFTs conducted within four weeks prior to randomization (e.g., collected as part of routine detoxification admission) will be acceptable. For participants whose induction onto their assigned study medication is delayed for longer than 2 weeks after randomization, LFTs and urine pregnancy should be repeated prior to start of study medication.

At screening, blood will be collected for HIV antibody, hepatitis C virus (HCV) antibody and hepatitis B surface antigen (HBsAG) and hepatitis B surface antibody (HBsAB) tests. These tests do not determine eligibility and will only be conducted on samples from participants who are randomized. Results of HIV antibody, hepatitis C virus (HCV) antibody and hepatitis B surface antigen (HBsAG) and hepatitis B surface antibody (HBsAB) tests conducted within four

weeks prior to randomization (e.g., collected as part of routine detoxification admission) will be acceptable.

For participants whose induction onto their assigned study medication occurs within 2 weeks of Day 0, LFTs will be repeated at week 4, week 12, and at the end-of-medication visit (if medication is stopped early) or at the end-of-treatment visit (week 24). For participants whose induction onto their assigned study medication occurs more than 2 weeks after day 0, LFTs will be repeated approximately 4 and 12 weeks following induction (a +/- 2 week window for post-induction LFTs is permitted), and at the end-of-medication visit (if medication is stopped early) or at the end-of-treatment visit (week 24). For participants who do not get inducted but continue on study, LFTs need not to be repeated at any of the planned visits with scheduled LFTs.

A laboratory that is accredited by the College of American Pathologists (CAP) or equivalent, and participates in the Clinical Laboratory Improvement Act of 1998 (CLIA) will perform these analyses. The laboratory will provide normal values and proof of lab certifications.

Changes in the liver function test values (alkaline phosphatase, ALT, AST, GGT and total bilirubin) over time and by treatment arm will be considered graphically. A listing of participants with elevated AST and ALT by treatment arm will be presented.

#### 7.4.1 Adverse Events (AEs) and Serious Adverse Events (SAEs)

At each medical management visit the study clinician will assess for AEs and SAEs by asking the study participant, "How have you been feeling since your last visit?" AEs and SAEs may also be spontaneously reported to study staff at any visit following consent. AEs and SAEs suggesting medical or psychiatric deterioration will be brought to the attention of a study clinician for further evaluation and management. Medical management visits will emphasize overdose risk and risk-management; any reported overdose will be recorded as an AE or SAE. AE and SAE reporting will be according to the reporting definitions and procedures outlined in the protocol and in accordance with applicable regulatory requirements.

For the purpose of this study, the following AE will not require reporting in the data system but will be captured in the source documentation as medically indicated:

Grade 1 (mild) unrelated adverse events

This would typically include mild physical events such as headache, cold, etc., that were considered not reasonably associated with the use of the study drug/intervention.

Events related to the injection of the study medication will be recorded on the Injection Site Abnormality (INA) form and will not be duplicate-reported on an AE form (See Section 7.4 for details on Injection Site examination summaries). Events related to withdrawal symptoms will be captured on the SOWS and HAM-D and will not be duplicate-reported on an AE form. Withdrawal symptoms not captured by the SOWS or HAM-D should be reported as an AE. Events captured on study specific forms (INA, SOWS, HAM-D) will not be recorded separately as an AE, unless they meet the SAE definition. Any of these events that meet the definition of an SAE will be reported on the AE/SAE form set. Any spontaneous reporting of withdrawal symptoms by the participant will be captured on AE form in the following situations: withdrawal symptoms reported at visits without scheduled specific structured questionnaires (SOWS, HAM-D); and withdrawal symptoms not listed in the specific structured questionnaires (SOWS, HAM-D) reported at any visit.

Adverse events (AEs), including serious adverse events (SAEs), will be summarized by body system and preferred term using MedDRA (The Medical Dictionary for Regulatory Activities) version 19.0 or higher. Adverse events will be presented in two ways: (1) the number and proportion of participants experiencing at least one incidence of each event will be presented overall and by treatment group. The incidence of adverse events and serious adverse events by

type will be compared between treatment arms using either Fisher's Exact mid-p-value or Chi-Square analysis as appropriate; and (2) a table displaying the total number of each event will be given overall and by treatment group. Listings of serious adverse events will be given, sorted by treatment, body system and preferred term. Detail in these listings will include severity, relationship to study drug, and action taken as available.

Treatment emergent AEs are defined as AEs occurring after participants have been inducted on study medication. Induction is defined as having had an injection if in the XR-NTX arm or having been dispensed medication if in the BUP-NX arm.

#### 7.5 Injection Site Examination

Appropriately qualified and trained medical personnel will examine the injection site on the next Medical Management visit following the XR-NTX administration. Participants will be asked to immediately report any injection site reactions to study staff for evaluation, monitoring, and possible referral, as needed. Injection site reactions should be documented on the Injection Site Abnormality Log. A detailed listing of injection site abnormalities will be provided.

#### 8.0 REFERENCES

Brooks AC, Comer SD, Sullivan MA, et al. Long-acting injectable versus oral naltrexone maintenance therapy with psychosocial intervention for heroin dependence: a quasi-experiment. J Clin Psychiatry. Oct 2010;71(10):1371-1378.

Carpenter KM, Jiang H, Sullivan MA, et al. Betting on change: modeling transitional probabilities to guide therapy development for opioid dependence. Psychol Addict Behav. Mar 2009;23(1):47-55.

Gail, M and Simon, R. Testing for Qualitative Interactions Between Treatment Effects and Patient Subsets. Biometrics. June 1985: 41: 361-372.

Mattick RP, Kimber J, Breen C, Davoli M. Buprenorphine maintenance versus placebo or methadone maintenance for opioid dependence. Cochrane Database Syst Rev. 2008(2):CD002207.

Nunes E, Hu M, Pavlicova M, Campbell A, Miele G, Hien D, Klein DF. Baseline matters: The importance of covariation for baseline severity in the analysis of clinical trials. Am J Drug Alcohol Abuse. Sep 2011;37(5):446-452.

Pocock SJ, Assmann SE, Enos LE, Kasten LE. Subgroup analysis, covariate adjustment and baseline comparisons in clinical trial reporting: current practice and problems. Stat Med. Oct 15 2002;21(19):2917-2930.

Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. Jul 2007;164(7):1035-1043.

Sullivan MA, Rothenberg JL, Vosburg SK, et al. Predictors of retention in naltrexone maintenance for opioid dependence: analysis of a stage I trial. Am J Addict. Mar-Apr 2006;15(2):150-159.

Trivedi MH, Wisniewski SR, Morris DW, et al. Concise Health Risk Tracking scale: a brief self-report and clinician rating of suicidal risk. J Clin Psychiatry. Jun 2011;72(6):757-64.





Figure 2: Randomization Status by CTP

Example figure provided.
CTN-0051: X:BOT Version 3.0 Statistical Analysis Plan April 27, 2017



Figure 3: Overall Expected vs. Actual Randomizations

Example figure provided.

Figure 4A: Early Randomizers Actual Randomizations

Similar Example Figure to Figure 3

Figure 5B: Late Randomizers Actual Randomizations

Similar Example Figure to Figure 3

| Table 1: Summary of Consents, Eligible Screens and Randomizations by CTP | | | | | |
|---|---|---|---|---|---|
| СТР | Number<br>of<br>Consents | Number<br>of<br>Eligible<br>Screens | Number<br>Randomized | Percent of<br>Consents<br>Randomized | Percent of<br>Eligible<br>Screens<br>Randomized |
| OV Maryhaven | | | | | |
| FL Gateway Community Services | | | | | |
| PA Tarzana Treatment Centers | | | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | | | | | |
| GNY Bellevue Hospital Center | | | | | |
| PNW ETS/RCKC | | | | | |
| MA Avery Road | | | | | |
| SW Turquoise Lodge Hospital | | | | | |
| Total | | | | | |

| | | Tab | ole 2: Summ | ary of Screen Fa | ilures by CTF | • | | | |
|---|---|---|---|---|---|---|---|---|---|
| | OV<br>Maryhaven | FL Gateway<br>Community<br>Services | PA Tarzana<br>Treatment<br>Centers | NEC Stanley<br>Street Treatment<br>and Resources<br>(SSTAR) | GNY Bellevue<br>Hospital<br>Center | PNW<br>ETS/RCKC | MA Avery<br>Road | SW<br>Turquoise<br>Lodge<br>Hospital | Total |
| Number of Consented | | | | | | | | | |
| Number of Screen Failures | | | | | | | | | |
| Eligibility Criteria Violated* (N (%)) | | | | | | | | | |
| 18 years of age or older | | | | | | | | | |
| Opioid use disorder | | | | | | | | | |
| Opioid use past 30 days | | | | | | | | | |
| Willing to accept random assignment | | | | | | | | | |
| Agrees to use birth control | | | | | | | | | |
| In good-enough health | | | | | | | | | |
| Able to provide written informed consent | | | | | | | | | |
| Able to speak<br>English/provide consent | | | | | | | | | |
| Severe medical, psychiatric, substance use condition | | | | | | | | | |
| Has LFTs greater than 5 times upper limit of normal | | | | | | | | | |
| Has suicidal or homicidal ideation | | | | | | | | | |
| Has allergy | | | | | | | | | |
| On methadone<br>maintenance | | | | | | | | | |
| Pain requiring opioid tx | | | | | | | | | |
| Pending legal action | | | | | | | | | |
| Pregnant/breastfeeding | | | | | | | | | |
| Inadequate body habitus | | | | | | | | | |

| | Table 2: Summary of Screen Failures by CTP | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | OV<br>Maryhaven | FL Gateway<br>Community<br>Services | PA Tarzana<br>Treatment<br>Centers | NEC Stanley<br>Street Treatment<br>and Resources<br>(SSTAR) | GNY Bellevue<br>Hospital<br>Center | PNW<br>ETS/RCKC | MA Avery<br>Road | SW<br>Turquoise<br>Lodge<br>Hospital | Total |
| Screening Visit Not<br>Completed | | | | | | | | | |
| Reasons for Not Completing the Screening Visit (N (%)) | | | | | | | | | |
| Participant dropped out of CTP | | | | | | | | | |
| Participant did not meet eligibility criteria | | | | | | | | | |
| Participant did not want research | | | | | | | | | |
| Other | | | | | | | | | |
| Number and Percentage of<br>Participants Eligible, but not<br>Randomized | | | | | | | | | |
| Reasons for Not Being<br>Randomized (N (%)) | | | | | | | | | |
| Participant dropped out of CTP | | | | | | | | | |
| Participant did not meet eligibility criteria | | | | | | | | | |
| Participant did not want research | | | | | | | | | |
| Other | | | | | | | | | |

<sup>\*</sup> Percentages are calculated based on the denominator of number of ineligibles and the sum may exceed 100% if multiple eligibility criteria are not met for potential participants.

| Table 3: Summary of the Timing of Randomization by CTP | | | |
|---|---|---|---|
| СТР | #<br>Randomized | # of Early<br>Randomizers <sup>1</sup> | # of Late<br>Randomizers <sup>1</sup> |
| OV Maryhaven | | | |
| FL Gateway Community Services | | | |
| PA Tarzana Treatment Centers | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | | | |
| GNY Bellevue Hospital Center | | | |
| PNW ETS/RCKC | | | |
| MA Avery Road | | | |
| SW Turquoise Lodge Hospital | | | |
| Total | | | |

<sup>&</sup>lt;sup>1</sup> Early randomizers are participants randomized within 72 hours following the last licit or illicit opioid use. Late randomizers are participants randomized greater than 72 hours following the last licit or illicit opioid use.

| | Tr | eatment Ar | m |
|---|---|---|---|
| | BUP-NX | XR-NTX | Total |
| Number of Randomized Participants | | | |
| Number Completing Week 24 visit - N (%) | | | |
| Number Completing Week 28 visit - N (%) | | | |
| Number of Study Completers <sup>1</sup> - N (%) | | | |
| Number of Early Terminations - N (%) | | | |
| Reasons for Early Termination | | | |
| Participant failed to return to clinic and unable to contact | | | |
| Participant terminated due to protocol deviation | | | |
| Participant terminated due to practical problems (no childcare, transportation, other) | | | |
| Participant moved from area | | | |
| Participant incarcerated | | | |
| Participant terminated due to AE/SAE | | | |
| Participant terminated for other clinical reasons | | | |
| Participant had a significant psychiatric risk (suicidal, homicidal, psychotic) | | | |
| Participant withdrew consent | | | |
| Participant deceased | | | |
| Participant terminated for other reason | | | |

<sup>&</sup>lt;sup>1</sup> Study completion is defined based on the Study Termination form and means that the subject completed the Week 36 visit.

| Table 5: Randomization by CTP and Stratification Factor | | | | |
|---|---|---|---|---|
| СТР | Opioid<br>Severity<br>Level <sup>1</sup> | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| OV Maryhaven | Low Severity | | | |
| | High<br>Severity | | | |
| FL Gateway Community Services | Low Severity | | | |
| | High<br>Severity | | | |
| PA Tarzana Treatment Centers | Low Severity | | | |
| | High<br>Severity | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | Low Severity | | | |
| | High<br>Severity | | | |
| GNY Bellevue Hospital Center | Low Severity | | | |
| | High<br>Severity | | | |
| PNW ETS/RCKC | Low Severity | | | |
| | High<br>Severity | | | |
| MA Avery Road | Low Severity | | | |
| | High<br>Severity | | | |
| SW Turquoise Lodge Hospital | Low Severity | | | |
| | High<br>Severity | | | |
| Total | Low Severity | | | |
| | High<br>Severity | | | |

| Table 5a: Randomization by CTP and Stratification Factor for Early Randomizers | | | | |
|---|---|---|---|---|
| СТР | Opioid<br>Severity<br>Level <sup>1</sup> | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| OV Maryhaven | Low Severity | | | |
| | High Severity | | | |
| FL Gateway Community Services | Low Severity | | | |
| | High Severity | | | |
| PA Tarzana Treatment Centers | Low Severity | | | |
| | High Severity | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | Low Severity | | | |
| | High Severity | | | |
| GNY Bellevue Hospital Center | Low Severity | | | |
| | High Severity | | | |
| PNW ETS/RCKC | Low Severity | | | |
| | High Severity | | | |
| MA Avery Road | Low Severity | | | |
| | High Severity | | | |
| SW Turquoise Lodge Hospital | Low Severity | | | |
| | High Severity | | | |
| Total | Low Severity | | | |
| | High Severity | | | |

<sup>&</sup>lt;sup>1</sup> To compute the opioid severity level, if the primary opioid of use in the last 7 days was not heroin or the route of administration is not IV-injection, then the participant is categorized in the low severity group. For IV heroin users where the quantity is not provided in bags but in dollars, bags are estimated as the dollar amount/10 rounded to the nearest integer.

| СТР | Opioid<br>severity<br>level <sup>1</sup> | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|
| OV Maryhaven | Low Severity | | | |
| | High<br>Severity | | | |
| FL Gateway Community Services | Low Severity | | | |
| | High<br>Severity | | | |
| PA Tarzana Treatment Centers | Low Severity | | | |
| | High<br>Severity | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | Low Severity | | | |
| | High<br>Severity | | | |
| GNY Bellevue Hospital Center | Low Severity | | | |
| | High<br>Severity | | | |
| PNW ETS/RCKC | Low Severity | | | |
| | High<br>Severity | | | |
| MA Avery Road | Low Severity | | | |
| | High<br>Severity | | | |
| SW Turquoise Lodge Hospital | Low Severity | | | |
| | High<br>Severity | | | |
| Total | Low Severity | | | |
| | High<br>Severity | | | |

<sup>&</sup>lt;sup>1</sup> Number of bags is assigned a 0 if the primary opioid of use in the last 7 days was not heroin or the route of administration is not IV-injection. For IV heroin users where the quantity is not provided in bags but in dollars, bags are estimated as the dollar amount/10 rounded to the nearest integer.

| Table 6: Summary of Study Medication I | iduction by Treatment Arm | | |
|---|---|---|---|
| | Т | reatment A | rm |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Induction Status | | | |
| Induction failure | | | |
| Inducted onto study medication | | | |
| Reasons for Induction Failure | | | |
| Participant could not tolerate detoxification | | | |
| Participant failed naloxone challenge | | | |
| Participant failed to provide a negative urine sample | | | |
| Participant left prior to induction | | | |
| Participant rejected treatment assignment | | | |
| Participant met criteria for relapse | | | |
| Participant reached end of induction window | | | |
| Time to Study Medication Induction (days) | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

| | _ | P-NX<br> =) | XR-NTX<br>(N=) | |
|---|---|---|---|---|
| | Inducted | Not Inducted | Inducted | Not Inducted |
| | N (%) | N (%) | N (%) | N (%) |
| Total | | | | |
| Randomization Timing Status | | | | |
| Early Randomizers | | | | |
| Late Randomizers | | | | |
| Opioid Severity Level <sup>1</sup> | | | | |
| Low Severity | | | | |
| High Severity | | | | |
| Randomization Timing Status by Opioid<br>Severity Level | | | | |
| Early Randomizers and Low Severity | | | | |
| Early Randomizers and High Severity | | | | |
| Late Randomizers and Low Severity | | | | |
| Late Randomizers and High Severity | | | | |
| Baseline Preference <sup>2</sup> | | | | |
| Preferred Neither Treatment | | | | |
| BUP-NX Preference | | | | |
| XR-NTX Preference | | | | |
| Preferred Either Treatment | | | | |

<sup>&</sup>lt;sup>1</sup> Number of bags is assigned a 0 if the primary opioid of use in the last 7 days was not heroin or the route of administration is not IV-injection. For IV heroin users where the quantity is not provided in bags but in dollars, bags are estimated as the dollar amount/10 rounded to the nearest integer.

<sup>&</sup>lt;sup>2</sup> Baseline preference is captured on the Motivation for Participating, Attitudes Regarding Study Medication form. The two questions to address preference are "I would prefer to receive Buprenorphine-Naloxone (Suboxone)" and "I would prefer to receive Naltrexone monthly injections" with responses to each on a 1 -5 scale of agreement with 1 indicating Strongly Disagree and 5 indicating Strongly Agree. If a participant indicates agreement or strong agreement, he/she will be deemed as having preferred that treatment. If the participant indicated agreement for both questions, he/she will be categorized as preferred either.

| | Т | reatment Aı | m |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Number of Early Medication Terminations - N (%) | | | |
| Reasons for Early Medication Termination | | | |
| Participant became pregnant | | | |
| Participant feels study treatment no longer necessary, not working | | | |
| Participant became incarcerated | | | |
| Participant withdrew consent | | | |
| Participant moved from area | | | |
| Participant deceased | | | |
| Participant met criteria for relapse | | | |
| Participant unable to tolerate side effects | | | |
| Participant continued to experience intolerable side effects after a dose reduction | | | |
| Contraindicated concomitant medication | | | |
| Participant refused, non-specific | | | |
| Participant left study and never returned | | | |
| Clinical deterioration: new onset of psychiatric or medical condition | | | |
| Physical illness or condition that precludes taking study medication | | | |
| Participant feels study treatment no longer necessary, cured | | | |
| Other | | | |

<sup>\*</sup>Note: Only participants inducted onto study medication are assessed for early medication termination.

| Table 9: Summary of Baseline Characteristics by Treatment Arm | | | |
|---|---|---|---|
| Characteristic | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Gender | | | |
| Missing | | | |
| Male | | | |
| Female | | | |
| Participant chose not to answer | | | |
| Age (Mean(Std)) | | | |
| Age | | | |
| Missing | | | |
| < 18 | | | |
| 18 - < 25 | | | |
| 25 - < 35 | | | |
| 35 - < 45 | | | |
| 45 - < 55 | | | |
| 55 - < 65 | | | |
| 65 - < 75 | | | |
| 75+ | | | |
| Ethnicity | | | |
| Not Hispanic or Latino | | | |
| Hispanic or Latino | | | |
| Missing | | | |
| Participant chose not to answer | | | |
| Race | | | |
| Missing | | | |
| American Indian or Alaska Native | | | |
| Asian | | | |
| Black or African American | | | |
| Native Hawaiian or Pacific Islander | | | |
| White | | | |
| Other | | | |
| Multiracial | | | |
| Unknown | | | |
| Participant chose not to answer | | | |

| Table 9: Summary of Baseline Characteristic | cs by Treatme | ent Arm | |
|---|---|---|---|
| Characteristic | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Education completed | | | |
| Less than high school diploma | | | |
| High school graduate | | | |
| GED or equivalent | | | |
| Some college, no degree | | | |
| Associate's degree: occupational, technical, or vocational program | | | |
| Associate's degree: academic program | | | |
| Bachelor's degree | | | |
| Master's degree | | | |
| Professional school degree | | | |
| Doctoral degree | | | |
| Don't know | | | |
| Refused | | | |
| Marital status <sup>1</sup> | | | |
| Married | | | |
| Widowed | | | |
| Divorced | | | |
| Separated | | | |
| Never married | | | |
| Living with partner | | | |
| Refused | | | |
| Don't know | | | |
| Employment | | | |
| Working now | | | |
| Only temporarily laid off, sick leave, or maternity leave | | | |
| Looking for work, unemployed | | | |
| Retired | | | |
| Disabled permanently or temporarily | | | |
| Keeping house | | | |
| Student | | | |
| Other | | | |

<sup>&</sup>lt;sup>1</sup> As defined on the DEM form.

| Table 10: Summary of Baseline Moderators by T | reatment | Arm | |
|---|---|---|---|
| | Т | reatment A | rm |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| IV Use | | | |
| Yes | | | |
| No | | | |
| Primary Opioid Used in the 7 Days Prior to Detox Admission | | | |
| Buprenorphine | | | |
| Opioid Analgesics | | | |
| Methadone | | | |
| Heroin | | | |
| Missing | | | |
| Cost per Day for Primary Opioid (dollars) | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Usual Living Arrangements (past 3 years) <sup>1</sup> | | | |
| With sexual partner and children | | | |
| With sexual partner alone | | | |
| With children alone | | | |
| With parents | | | |
| With family | | | |
| With friends | | | |
| Alone | | | |
| Controlled environment | | | |
| No stable arrangements | | | |
| Not answered | | | |
| Any Friends and/or Family Members with Alcohol Problems | | | |
| Yes | | | |
| No | | | |
| Any Friends and/or Family Members that Use Heroin and/or Other Illicit Opioids | | | |
| Yes | | | |
| No | | | |
| Any Friends and/or Family Members that Use Illicit Drugs and/or Non-prescribed Drugs | | | |
| Yes | | | |
| No | | | |
| If I receive BUP-NX I am sure that I will take it every day for the next 6 months. | | | |
| Strongly disagree | | | |

| | Т | reatment A | rm |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Disagree | , | , , | |
| Neutral | | | |
| Agree | | | |
| Strongly Agree | | | |
| If I receive XR-NTX I am sure that I will get an injection every month for the next 6 months. | | | |
| Strongly disagree | | | |
| Disagree | | | |
| Neutral | | | |
| Agree | | | |
| Strongly Agree | | | |
| Ever Heroin Use (Lifetime use based on ASI collected at Baseline) | | | |
| Yes | | | |
| No | | | |
| Current Heroin Use (Past 30 day use based on ASI collected at Baseline) | | | |
| Yes | | | |
| No | | | |
| Ever Prescription Opioid Use (Lifetime use based on ASI collected at Baseline) | | | |
| Yes | | | |
| No | | | |
| Current Prescription Opioid Use (Past 30 day use based on ASI collected at Baseline) | | | |
| Yes | | | |
| No | | | |
| Current Age | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Age at Onset of Any Opioid Use | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max Duration of Opioid Use (Current age minus Age at onset of any opioids based on Baseline ASI) | | | |
| Mean | | | |
| SD | | | |

| | Т | reatment A | rm |
|---|---|---|---|
| | BUP-NX | XR-NTX | Tota |
| | (N=) | (N=) | (N=) |
| Median | | | |
| Min | | | |
| Max | | | |
| First Treatment Status <sup>2</sup> | | | |
| Yes | | | |
| No | | | |
| Past Treatment Successful <sup>3</sup> | | | |
| Yes | | | |
| No | | | |
| Any Stimulants Use | | | |
| Yes | | | |
| No | | | |
| Any Sedatives Use | | | |
| Yes | | | |
| No | | | |
| Any Alcohol Heavy Drinking Days⁴ | | | |
| Yes | | | |
| No | | | |
| Any Cannabis Use | | | |
| Yes | | | |
| No | | | |
| HAM-D Score (Baseline) | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| ASI Psychiatric Domain Composite Score (Baseline) | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Any History of Psychiatric Disorders from Medical History <sup>5</sup> | | | |
| Yes | | | |
| No | | | |
| Discomfort Level of Past Opioid Withdrawal (Scale of 0 to 10) | | | |

| Table 10: Summary of Bas | eline Moderators by Treatment Arm | |
|--------------------------|-----------------------------------|-------------|
| | Treatment Arm | |
| | | otal<br>N=) |
| Mean | | |
| SD | | |
| Median | | |
| Min | | |
| Max | | |
| SOWS Score at Baseline | | |
| Mean | | |
| SD | | |
| Median | | |
| Min | | |
| Max | | |

<sup>&</sup>lt;sup>1</sup> Based on the ASI Family/Social Relationships section.

<sup>&</sup>lt;sup>2</sup> The first treatment status is defined based on the participants response to the Opiate Treatment History provided on the MHX form. If the subject indicated No for the history of any treatments, then this is his/her first episode of treatment.

<sup>&</sup>lt;sup>3</sup> Past treatment successful is only tabulated for those who were previously treated.

Heavy Drinking days is defined as a day that a man has 5 or more drinks or a woman has 4 or more drinks.

The following psychiatric disorders are collected on the Medical History: Anxiety or panic disorder, Attention Deficit Hyperactivity Disorder, Bipolar Disorder, Major Depressive Disorder, Schizophrenia, Suicidal ideation, Suicidal behavior, Homicidal ideation, Homicidal behavior, Violent behavior, Psychotic episodes, or other psychiatric disorder. If the subject responded Yes to any of those psychiatric disorders, he/she is categorized as Yes to having had a psychiatric disorder.

| | Table 11: Summary of Treatment Exposure* by Treatment Arm | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| СТР | Participants<br>Randomized<br>to BUP-NX | Expected Days<br>(Buprenorphine<br>Arm) | Actual Days<br>Taken<br>(Buprenorphine<br>Arm) | Buprenorphine<br>Exposure<br>Percentage | Participa<br>nts<br>Randomiz<br>ed to XR-<br>NTX | Expected<br>Vivitrol<br>Injections | Actual<br>Vivitrol<br>Injections | Vivitrol<br>Exposure<br>Percentage |
| OV Maryhaven | | | | | | | | |
| FL Gateway Community Services | | | | | | | | |
| PA Tarzana Treatment Centers | | | | | | | | |
| NEC Stanley Street Treatment and Resources | | | | | | | | |
| GNY Bellevue Hospital Center | | | | | | | | |
| PNW ETS/RCKC | | | | | | | | |
| MA Avery Road | | | | | | | | |
| SW Turquoise Lodge Hospital | | | | | | | | |
| Overall | | | | | | | | |

<sup>\*</sup>Treatment Exposure is calculated only for participants who have been inducted onto study medication.

The time period for treatment exposure begins at induction and ends at the onset of the relapse event or at the end of the study treatment period, whichever comes first.

| Table | Table 12: Summary of Vivitrol Injections and Injection Intervals by CTP | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | OV<br>Maryhaven | FL Gateway<br>Community<br>Services | PA Tarzana<br>Treatment<br>Centers | NEC<br>Stanley<br>Street<br>Treatment<br>and<br>Resources<br>(SSTAR) | GNY<br>Bellevue<br>Hospital<br>Center | PNW<br>ETS/RCKC | MA Avery<br>Road | SW<br>Turquoise<br>Lodge<br>Hospital | Total |
| Number of Participants Randomized to Vivitrol | | | | | | | | | |
| Number of Injections | | | | | | | | | |
| 1 | | | | | | | | | |
| 2 | | | | | | | | | |
| 3 | | | | | | | | | |
| 4 | | | | | | | | | |
| 5 | | | | | | | | | |
| 6 | | | | | | | | | |
| 7 | | | | | | | | | |
| Injection Intervals (days) <sup>1</sup> | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Injection intervals are defined as time between two consecutive injections. To have an injection interval, participants must have at least two injections. Participants with more than two injections will have multiple injection intervals included.

| Tak | Table 13: Summary of BUP-NX Prescribed Daily Dose by CTP | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | OV<br>Maryhaven | FL Gateway<br>Community<br>Services | PA Tarzana<br>Treatment<br>Centers | NEC<br>Stanley<br>Street<br>Treatment<br>and<br>Resources<br>(SSTAR) | GNY<br>Bellevue<br>Hospital<br>Center | PNW<br>ETS/RCKC | MA Avery<br>Road | SW<br>Turquoise<br>Lodge<br>Hospital | Total |
| Number of Participants Randomized to BUP-NX | | | | | | | | | |
| Maximum Prescribed Daily Dose Across all Visits | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| Minimum Prescribed Daily Dose Across all Visits | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |

Figure 6: Participant-level Prescribed Daily Dose of Buprenorphine



Example figure provided.

| Table 14: Availability of Primary Outcome by Treatment Arm (Day 21 – Day 167*) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment<br>Arm | Participants<br>Randomized | Number<br>of UDS<br>Collected | Number<br>of UDS<br>Expected | Percentage<br>of UDS<br>Collected | Number<br>of TLFB<br>Days<br>Collected | Number<br>of TLFB<br>Days<br>Expected | Percentage<br>of TLFB<br>Days<br>Collected | Availability<br>of Primary<br>Outcome** |
| BUP-NX | | | | | | | | |
| XR-NTX | | | | | | | | |
| Total | | | | | | | | |

<sup>\*</sup>Day 167 or the last day of the relapse event, whichever occurs first, for participants who have been inducted onto study medication.

<sup>\*\*</sup>The Availability of Primary Outcome is the average of the percentage of expected TLFB days collected and percentage of expected UDS collected.

| | Treatment Arm | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Relapse Status <sup>1</sup> | | | |
| Yes | | | |
| No | | | |
| Time to Relapse <sup>2</sup> (days) | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Percentage of Opioid Use Days based on TLFB <sup>3</sup> (Day 0-21 post-randomization) (%) | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| UDS Result at Randomization (Day 0) | | | |
| Positive for non-prescribed Opioids | | | |
| Negative for non-prescribed Opioids | | | |
| Missing | | | |
| UDS Result at Week 1 (Day 3-12) | | | |
| Positive for non-prescribed Opioids | | | |
| Negative for non-prescribed Opioids | | | |
| Missing | | | |
| UDS Result at Week 2 (Day 10-16) | | | |
| Positive for non-prescribed Opioids | | | |
| Negative for non-prescribed Opioids | | | |
| Missing | | | |
| UDS Result at Week 3 (Day 17-23) | | | |
| Positive for non-prescribed Opioids | | | |
| Negative for non-prescribed Opioids | | | |
| Missing | | | |

<sup>&</sup>lt;sup>1</sup> A participant is defined as not having relapsed if by the Week 24 visit, the participant did not meet any of the relapse criteria. <sup>2</sup> Time to relapse summary statistics are only summarized for subjects who met the relapse criteria. <sup>3</sup> Participants do not provide TLFB data while in detox.

Figure 5A: TLFB and UDS for Day 0 to Day 21Figure 5A: UDS for Day 0 to Day 21-Treatment=BUP-NX

Figure 5B: UDS for Day 0 to Day 21- Treatment=XR-NTX

Figure 5C: TLFB for Day 0 to Day 21- Treatment=BUP-NX

Figure 5D: TLFB for Day 0 to Day 21- Treatment=XR-NTX



Separate figures will be generated for TLFB and UDS and additionally separate for each treatment arm. Each row in the figure would correspond with a participants TLFB and UDS results only from Day 0 to Day 21. The legend would indicate that the green vertical dashes indicate no illicit opioid use on TLFB whereas the yellow vertical dashes indicate illicit opioid use. The red +, - and o values indicate UDS results of positive for non-protocol defined opioids, negative for non-protocol defined opioids and missing UDS results respectively. The figure colors will be modified to accommodate color blind readers.

Figure 6: Kaplan-Meier Plots of Time to Relapse by Treatment Arm

Example Kaplan-Meier figure provided below.



The x-axis for the Time to Relapse Kaplan-Meier Plots will be measured in days. Separate curves on the same plot will be defined as the treatment arms. Censored observations will be represented using a + sign.

| Table 16: Summary of Primary Outcome (Time to Relapse <sup>1</sup> ) for Groups of Interest | | | | | | |
|---|---|---|---|---|---|---|
| | | BUP-NX<br>(N=) | | | XR-NTX<br>(N=) | |
| | N | Mean<br>(STD) | Median<br>(Min, Max) | N | Mean<br>(STD) | Median<br>(Min, Max) |
| Randomization Timing Status | | | | | | |
| Early Randomizers | | | | | | |
| Late Randomizers | | | | | | |
| Opioid Severity Level | | | | | | |
| Low Severity | | | | | | |
| High Severity | | | | | | |
| Randomization Timing Status by Opioid Severity Level | | | | | | |
| Early Randomizers and Low Severity | | | | | | |
| Early Randomizers and High Severity | | | | | | |
| Late Randomizers and Low Severity | | | | | | |
| Late Randomizers and High Severity | | | | | | |
| Inducted onto Study Medication | | | | | | |
| Baseline Preference <sup>2</sup> | | | | | | |
| Preferred Neither Treatment | | | | | | |
| BUP-NX Preference | | | | | | |
| XR-NTX Preference | | | | | | |
| Preferred Either Treatment | | | | | | |
| Baseline Motivation <sup>3</sup> | | | | | | |
| Motivated for Neither Treatment | | | | | | |
| BUP-NX Motivated | | | | | | |
| XR-NTX Motivated | | | | | | |
| Motivated for Both Treatments | | | | | | |

<sup>&</sup>lt;sup>1</sup> Time to relapse summary statistics are only summarized for subjects who met the relapse criteria.

<sup>&</sup>lt;sup>2</sup> Baseline preference is captured on the Motivation for Participating, Attitudes Regarding Study Medication form. The two questions to address preference are "I would prefer to receive Buprenorphine-Naloxone (Suboxone)" and "I would prefer to receive Naltrexone monthly injections" with responses to each on a 1 -5 scale of agreement with 1 indicating Strongly Disagree and 5 indicating Strongly Agree. If a participant indicates agreement or strong agreement, he/she is deemed as having preferred that treatment. If the participant indicated agreement for both questions, he/she is categorized as preferred either.

<sup>&</sup>lt;sup>3</sup>Baseline motivation is captured on the Motivation for Participating, Attitudes Regarding Study Medication form. The two questions to address motivation are "If I receive Buprenorphine-Naloxone (Suboxone) I am sure that I will take it every day for the next 6 months." and "If I receive Naltrexone I am sure that I will get an injection every month for the next 6 months" with responses to each on a 1-5 scale of agreement with 1 indicating Strongly Disagree and 5 indicating Strongly Agree. If a participant indicates agreement or strong agreement, he/she is deemed as being motivated. If the participant indicated agreement for both questions, he/she is categorized as Motivated for Both Treatments.

## Figure 7: Kaplan-Meier Plots of Time to Relapse by Randomization Timing Status and Treatment Arm

Example Kaplan-Meier figure provided in Figure 6.

Four separate curves for each treatment arm and randomization timing status will be plotted on one figure.

## Figure 8: Kaplan-Meier Plots of Time to Relapse by Opioid Severity Level and Treatment Arm

Example Kaplan-Meier figure provided in Figure 6.

Four separate curves for each treatment arm and opioid severity level will be plotted on one figure.

## Figure 9: Kaplan-Meier Plots of Time to Relapse by Randomization Timing, Opioid Severity Level and Treatment Arm

Example Kaplan-Meier figure provided in Figure 6.

Four separate curves for each treatment arm, opioid severity level and randomization timing will be plotted on one figure.

| | Table | 17: Summ | ary of Prim | nary Outcor | ne (Rela | ose) by C | ГР | | |
|---|---|---|---|---|---|---|---|---|---|
| | OV<br>Maryhaven<br>(N=) | FL<br>Gateway<br>Community<br>Services<br>(N=) | PA Tarzana<br>Treatment<br>Centers<br>(N=) | NEC Stanley Street Treatment and Resources (SSTAR) (N=) | GNY<br>Bellevue<br>Hospital<br>Center<br>(N=) | PNW<br>ETS/RCKC<br>(N=) | MA Avery<br>Road<br>(N=) | SW<br>Turquoise<br>Lodge<br>Hospital<br>(N=) | Total<br>(N=) |
| Relapse Status | | | | | | | | | |
| Yes | | | | | | | | | |
| No | | | | | | | | | |
| Time to Relapse <sup>1</sup> (days) | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| Percentage of Opioid<br>Use Days based on<br>TLFB <sup>2</sup> (Day 0-21 post-<br>randomization) (%) | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| UDS Result at<br>Randomization (Day 0) | | | | | | | | | |
| Positive for non-<br>prescribed Opioids | | | | | | | | | |
| Negative for non-<br>prescribed Opioids Missing | | | | | | | | | |
| UDS Result at Week 1<br>(Day 3-12) | | | | | | | | | |
| Positive for non-<br>prescribed Opioids | | | | | | | | | |
| Negative for non-<br>prescribed Opioids | | | | | | | | | |
| Missing | | | | | | | | | |
| UDS Result at Week 2<br>(Day 10-16) | | | | | | | | | |
| Positive for non-<br>prescribed Opioids | | | | | | | | | |

| | OV<br>Maryhaven<br>(N=) | FL<br>Gateway<br>Community<br>Services<br>(N=) | PA Tarzana<br>Treatment<br>Centers<br>(N=) | NEC Stanley Street Treatment and Resources (SSTAR) (N=) | GNY<br>Bellevue<br>Hospital<br>Center<br>(N=) | PNW<br>ETS/RCKC<br>(N=) | MA Avery | SW<br>Turquoise<br>Lodge<br>Hospital<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|---|---|---|
| Negative for non-<br>prescribed Opioids | | | | | | | | | |
| Missing | | | | | | | | | |
| UDS Result at Week 3<br>(Day 17-23) | | | | | | | | | |
| Positive for non-<br>prescribed Opioids | | | | | | | | | |
| Negative for non-<br>prescribed Opioids | | | | | | | | | |
| Missing | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Time to relapse summary statistics are only summarized for subjects who met the relapse criteria. <sup>2</sup> Participants do not provide TLFB data while in detox.

| Table 18: Summary of Relapse Status <sup>1</sup> for the Groups of Interest | | | | |
|---|---|---|---|---|
| | | P-NX<br>I=) | XR-NTX<br>(N=) | |
| | Relapsed | Not Relapsed | Relapsed | Not Relapsed |
| | N (%) | N (%) | N (%) | N (%) |
| Total | | | | |
| Randomization Timing Status | | | | |
| Early Randomizers | | | | |
| Late Randomizers | | | | |
| Opioid Severity Level | | | | |
| Low Severity | | | | |
| High Severity | | | | |
| Randomization Timing Status by Opioid Severity Level | | | | |
| Early Randomizers and Low Severity | | | | |
| Early Randomizers and High Severity | | | | |
| Late Randomizers and Low Severity | | | | |
| Late Randomizers and High Severity | | | | |
| Inducted onto Study Medication | | | | |

<sup>&</sup>lt;sup>1</sup> A participant is defined as not having relapsed if by the Week 24 visit, the participant did not meet any of the relapse criteria.

| Table 19: Summary of Percent Days of Illicit Opioid Use <sup>1</sup> for Groups of Interest | | | | | | |
|---|---|---|---|---|---|---|
| | BUP-NX<br>(N=) | | | XR-NTX<br>(N=) | | |
| | N | Mean<br>(STD) | Median<br>(Min, Max) | N | Mean (STD) | Median<br>(Min, Max) |
| Randomization Timing Status | | | | | | |
| Early Randomizers | | | | | | |
| Late Randomizers | | | | | | |
| Opioid Severity Level | | | | | | |
| Low Severity | | | | | | |
| High Severity | | | | | | |
| Randomization Timing Status by Opioid Severity Level | | | | | | |
| Early Randomizers and Low Severity | | | | | | |
| Early Randomizers and High Severity | | | | | | |
| Late Randomizers and Low Severity | | | | | | |
| Late Randomizers and High Severity | | | | | | |
| Inducted onto Study Medication | | | | | | |

<sup>&</sup>lt;sup>1</sup> Percent days of illicit opioid use is calculated based on TLFB (only illicit use is provided) starting on Day 21 up until the day of relapse and is calculated as the number of opioid use divided by the total number of days in that time frame. Note, if the subject relapses immediately on Day 21, the percent days of opioid use is 100%. Missing TLFB days are defined as opioid use days.

| Table 20: Summary of Abstinent Days <sup>1</sup> for Groups of Interest | | | | | | |
|---|---|---|---|---|---|---|
| | BUP-NX<br>(N=) | | | | XR-NTX | |
| | | | | (N=) | | |
| | N | Mean<br>(STD) | Median<br>(Min, Max) | N | Mean (STD) | Median<br>(Min, Max) |
| Randomization Timing Status | | | | | | |
| Early Randomizers | | | | | | |
| Late Randomizers | | | | | | |
| Opioid Severity Level | | | | | | |
| Low Severity | | | | | | |
| High Severity | | | | | | |
| Randomization Timing Status by Opioid Severity Level | | | | | | |
| Early Randomizers and Low Severity | | | | | | |
| Early Randomizers and High Severity | | | | | | |
| Late Randomizers and Low Severity | | | | | | |
| Late Randomizers and High Severity | | | | | | |
| Inducted onto Study Medication | | | | | | |

<sup>&</sup>lt;sup>1</sup> Abstinent days are calculated based on TLFB starting on Day 21 up until the day of relapse and will be calculated as the number of days where opioids were not used. Missing TLFB days are defined as non-abstinent days.

| Table 21: Summary of Number of Visits 'Present and Clean' for Groups of Interest | | | | | | |
|---|---|---|---|---|---|---|
| | BUP-NX<br>(N=) | | | XR-NTX<br>(N=) | | |
| | N | Mean<br>(STD) | Median<br>(Min, Max) | N | Mean (STD) | Median<br>(Min, Max) |
| Randomization Timing Status | | | | | | |
| Early Randomizers | | | | | | |
| Late Randomizers | | | | | | |
| Opioid Severity Level | | | | | | |
| Low Severity | | | | | | |
| High Severity | | | | | | |
| Randomization Timing Status by Opioid Severity Level | | | | | | |
| Early Randomizers and Low Severity | | | | | | |
| Early Randomizers and High Severity | | | | | | |
| Late Randomizers and Low Severity | | | | | | |
| Late Randomizers and High Severity | | | | | | |
| Inducted onto Study Medication | | | | | | |

<sup>&</sup>lt;sup>1</sup> Number of Visits 'Present and Clean" is based on the UDS results evaluated starting at Day 21 and up until the point of relapse. A UDS result which is within temperature range and deemed to be unadulterated and is not positive for non-protocol prescribed opioids is categorized as present and clean. A complete number of UDS results 'Present and Clean" is defined for each participant.
| | BUP-<br>(N= | | X | R-NTX<br>(N=) |
|---|---|---|---|---|
| | Completed 24<br>Weeks of<br>Treatment<br>N (%) | Didn't<br>Complete 24<br>Weeks of<br>Treatment<br>N (%) | Completed 24<br>Weeks of<br>Treatment<br>N (%) | Didn't Complete 24<br>Weeks of Treatment<br>N (%) |
| Total | | | | |
| Randomization Timing Status | | | | |
| Early Randomizers | | | | |
| Late Randomizers | | | | |
| Opioid Severity Level <sup>1</sup> | | | | |
| Low Severity | | | | |
| High Severity | | | | |
| Randomization Timing Status by Opioid Severity Level | | | | |
| Early Randomizers and Low Severity | | | | |
| Early Randomizers and High Severity | | | | |
| Late Randomizers and Low Severity | | | | |
| Late Randomizers and High Severity | | | | |
| Baseline Preference <sup>2</sup> | | | | |
| Preferred Neither Treatment | | | | |
| BUP-NX Preference | | | | |
| XR-NTX Preference | | | | |
| Preferred Either Treatment | | | | |
| Inducted onto Study Medication | | | | |

<sup>&</sup>lt;sup>1</sup> A participant is defined as completing 24 weeks of treatment if he/she received XR-NTX in Week 20-24 or was dispensed BUP-NX during Week 20-24.

| | | | | Та | ble 23: | Sumi | mary o | f Trails | A and | B by | Treatm | ent A | rm | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Treatme | nt Arm | | | | | | | | |
| | | | BUP<br>(N | | | | | | XR-I<br>(N: | | | | | | To<br>(N | | | |
| | Week<br>0 | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | EOT | Week<br>0 | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | EOT | Week<br>0 | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | EOT |
| Trails A | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | | | | | |
| Trails B | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | | | | | |

CTN-0051: X:BOT Version 3.0 Statistical Analysis Plan April 27, 2017



Figure 10: Boxplots of Trails A by Treatment Arm

Example figure provided.

Figure 11: Boxplots of Trails B by Treatment Arm

| | | Та | ble 24 | Sum | mary o | of Str | oop C | olor ar | nd Wo | rd Sco | res by | / Trea | atment | Arm | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Treatme | ent Arm | | | | | | | | |
| | | | BUP<br>(N | | | | | | XR-I<br>(N | | | | | | To: | | | |
| | Week<br>0 | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | EOT | Week<br>0 | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | EOT | Week<br>0 | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | EOT |
| Word Score | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | | | | | |
| Color Score | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | | | | | |
| Color-Word Score | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | | | | | |

Version 3.0 April 27, 2017

## Figure 12: Boxplots of Stroop Word Score by Treatment Arm

See example box plot figure provided above.

## Figure 13: Boxplots of Stroop Color Score by Treatment Arm

See example box plot figure provided above.

## Figure 14: Boxplots of Stroop Color-Word Score by Treatment Arm

See example figure provided above.

| | | Treatment Arm | |
|----------------------|----------------|----------------|---------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| HAM-D Score – Week 0 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 1 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 2 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 3 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 4 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

| | | Treatment Arm | |
|-----------------------|----------------|----------------|---------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| HAM-D Score – Week 8 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 12 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 16 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 20 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| HAM-D Score – Week 24 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

CTN-0051: X:BOT Version 3.0 Statistical Analysis Plan April 27, 2017

Figure 15: Boxplots of HAM-D Score by Treatment Arm

| | | Treatment Arm | |
|---------------------|----------------|----------------|--------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Tota<br>(N=) |
| SOWS Score – Week 0 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 1 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 2 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 3 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 4 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 8 | | | |
| N | | | |

| | | Treatment Arm | |
|----------------------|----------------|----------------|--------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Tota<br>(N=) |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 12 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 16 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 20 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| SOWS Score – Week 24 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

Figure 16: Boxplots of SOWS Score by Treatment Arm

| | | Treatment Arm | |
|--------------------|----------------|----------------|---------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| VAS Score – Week 0 | , , | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 1 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 2 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 3 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 4 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 5 | | | |
| N | | | |
| Mean | | | |
| SD | | | |

| | | Treatment Arm | |
|---------------------|----------------|----------------|--------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Tota<br>(N=) |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 6 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 7 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Max | | | |
| VAS Score – Week 8 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 9 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 10 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

| | | Treatment Arm | |
|---------------------|----------------|----------------|---------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| VAS Score – Week 11 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 12 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 13 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 14 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 15 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 16 | | | |
| N | | | |
| Mean | | | |
| SD | | | |

| | | Treatment Arm | |
|---------------------|----------------|----------------|---------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 17 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Max | | | |
| VAS Score – Week 18 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 19 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 20 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 21 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

| | | Treatment Arm | |
|---------------------|----------------|----------------|---------------|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| VAS Score – Week 22 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 23 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| VAS Score – Week 24 | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

Figure 17: Boxplots of VAS Score by Treatment Arm

| Table 28: Summary of Self-Reported Alcohol Use by Treatment Arm | | | |
|---|---|---|---|
| | Treatment Arm | | |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Week 0 | , , | | |
| Alcohol Use in the Past 30 Days – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 1 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 2 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 3 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |

| | Treatment Arm | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 4 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days¹ – N (%) | | | |
| Week 5 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 6 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days¹ – N (%) | | | |
| Week 7 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |

| | | Treatment Arm | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 8 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days¹ – N (%) | | | |
| Week 9 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 10 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 11 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |

| | | <b>Treatment Arm</b> | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 12 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 13 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 14 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 15 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |

| Table 28: Summary of Self-Reported Alcohol Use by Treatment Arm | | | |
|---|---|---|---|
| | | Treatment Arm | |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 16 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 17 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 18 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 19 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |

| | Treatment Arm | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 20 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 21 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 22 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 23 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |

| | | <b>Treatment Arm</b> | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |
| Week 24 | | | |
| Alcohol Use Within Visit Window – N (%) | | | |
| Drinks per Day | | | |
| N | | | |
| Mean | | | |
| SD | | | |
| Median | | | |
| Min | | | |
| Max | | | |
| Heavy Drinking Days <sup>1</sup> – N (%) | | | |

<sup>&</sup>lt;sup>1</sup>A heavy drinking day is defined as 4 or more drinks for females and 5 or more for males.

| Table 29: Summary of Self-Reported Other Drug Use by Treatment Arm | | | |
|---|---|---|---|
| | Treatment Arm | | |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Week 0 | , , | , , | , , |
| Number of Available Participants | | | |
| Any Substance Use in the Past 30 Days – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 1 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 2 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 3 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 4 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 5 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 6 | | | |
| Number of Participants Available | | | |

| Table 29: Summary of Self-Reported Other Drug Use by Treatment Arm | | | |
|---|---|---|---|
| | Treatment Arm | | |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 7 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 8 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 9 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 10 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 11 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 12 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| · | | | <u> </u> |

| Table 29: Summary of Self-Reported Other Drug Use by Treatment Arm | | | |
|---|---|---|---|
| | Treatment Arm | | |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 13 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 14 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 15 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 16 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 17 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 18 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |

| | | Treatment Arm | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Week 19 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 20 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 21 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 22 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 23 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |
| Week 24 | | | |
| Number of Participants Available | | | |
| Any Substance Use Within Visit Window – N (%) | | | |
| Cannabis Use – N (%) | | | |
| Cocaine Use – N (%) | | | |
| Stimulant Use – N (%) | | | |

| | Treatment Arm | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Week 0 | , , | , , | , |
| Cigarettes per Day in Past 30 Days – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 1 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 2 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 3 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 4 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 5 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 6 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |

| T | -Reported Tobacco Use by Treatment Arm Treatment Arm | | |
|---|---|---|---|
| | DUD NY | | |
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| 11-20 | , , | , , | , , |
| 21-30 | | | |
| 31 or more | | | |
| Week 7 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 8 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 9 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 10 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 11 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 12 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |

| | | Treatment Arm | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Week 13 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 14 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 15 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 16 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 17 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 18 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 19 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |

| | | <b>Treatment Arm</b> | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 20 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 21 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 22 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 23 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |
| Week 24 | | | |
| Cigarettes per Day Within Visit Window – N (%) | | | |
| 10 or less | | | |
| 11-20 | | | |
| 21-30 | | | |
| 31 or more | | | |

| Table 31: Summary of Problems Related to Drug Abuse by Treatment Arm | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment Arm | | | | | | | | |
| | BUP-NX<br>(N=) | | | | XR-NTX<br>(N=) | Total<br>(N=) | | | |
| | Week 0 | Week<br>24 | Week<br>36 | Week 0 | Week<br>24 | Week<br>36 | Week<br>0 | Week<br>24 | Week<br>36 |
| ASI-Lite: Drug/Alcohol Use<br>Composite Score | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| ASI-Lite: Family/Social Relationships<br>Composite Score | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| ASI-Lite: General Information<br>Composite Score | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| ASI-Lite: Legal Status Composite<br>Score | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| ASI-Lite: Medical Status Composite<br>Score | | | | | | | | | |
| N | | | | | 1 | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| L | | | <u> </u> | <u> </u> | | | l | | l |

| Table 31: Summary of Problems Related to Drug Abuse by Treatment Arm | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment Arm | | | | | | | | |
| | BUP-NX<br>(N=) | | | XR-NTX<br>(N=) | | | Total<br>(N=) | | |
| | Week 0 | Week<br>24 | Week<br>36 | Week 0 | Week<br>24 | Week<br>36 | Week<br>0 | Week<br>24 | Week<br>36 |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| ASI-Lite: Psychiatric Status<br>Composite Score | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| EuroQoL Questionnaire Composite<br>Score | | | | | | | | | |
| N | | | | | | | | | |
| Mean | | | | | | | | | |
| SD | | | | | | | | | |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |

| Table 32: Summary of HIV Risk by Treatment Arm | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Treatment Arm | | | | | | | | | | |
| | BUP-NX<br>(N=) | | | | XR-NTX<br>(N=) | | | | Total<br>(N=) | | | |
| | Week 0 | Week 12 | Week 24 | Week<br>36 | Week 0 | Week 12 | Week<br>24 | Week 36 | Week 0 | Week 12 | Week 24 | Week 36 |
| Number of Times Participant had<br>Penetrative Sex (vaginal or anal<br>sex) in the Past 30 Days | | | | | | | | | | | | |
| N | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | |
| SD | | | | | | | | | | | | |
| Median | | | | | | | | | | | | |
| Min | | | | | | | | | | | | |
| Max | | | | | | | | | | | | |
| Number of Times Participant had<br>Penetrative Sex (vaginal or anal<br>sex) without a Condom in the<br>Past 30 Days | | | | | | | | | | | | |
| N | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | |
| SD | | | | | | | | | | | | |
| Median | | | | | | | | | | | | |
| Min | | | | | | | | | | | | |
| Max | | | | | | | | | | | | |
| | BUP-NX | XR-NTX | Total |
|---|---|---|---|
| N 1 (D (C) 1 (H T 1 (E) 1 (A) E 1 | (N=) | (N=) | (N=) |
| Number of Participants with Treatment Emergent Adverse Events | | | |
| Number of Treatment Emergent Adverse Events | | | |
| Severity of Treatment Emergent Adverse Event | | | |
| Grade 1-Mild | | | |
| Grade 2-Moderate | | | |
| Grade 3-Severe | | | |
| Relationship of Treatment Emergent Adverse Event | | | |
| Not Related | | | |
| Related | | | |

<sup>\*</sup>Note: Treatment emergence is defined as any adverse event that occurred after the study day of induction for those participants inducted onto study medication.

| Table 34: Summary of Treatment Emergent* Serious Adverse Events by Treatment Arm | | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Number of Participants Inducted | | | |
| Number of Participants with a Treatment Emergent Serious Adverse Event | | | |
| Number of Treatment Emergent Serious Adverse Events | | | |
| Type of Treatment Emergent Serious Adverse Event | | | |
| Death | | | |
| Life-threatening event | | | |
| Inpatient admission to hospital or prolongation of existing hospitalization | | | |
| Persistent or significant incapacity | | | |
| Congenital anomaly or birth defect | | | |
| Important medical event that required intervention to prevent any of the above | | | |
| Severity of Treatment Emergent Serious Adverse Event | | | |
| Grade 1-Mild | | | |
| Grade 2-Moderate | | | |
| Grade 3-Severe | | | |
| Relationship of Treatment Emergent Serious Adverse Event | | | |
| Not Related | | | |
| Related | | | |

<sup>\*</sup>Note: Treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.

| System Organ Class/ Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Participants with at least one treatment emergent adverse event | | | |
| Gastrointestinal disorders | | | |
| Constipation | | | |
| Vomiting | | | |
| Diarrhoea | | | |
| Nausea | | | |
| Toothache | | | |
| Abdominal pain upper | | | |
| Abdominal pain | | | |
| Glossitis | | | |
| Oral mucosal erythema | | | |
| Abdominal discomfort | | | |
| Glossodynia | | | |
| Gingival swelling | | | |
| Dyspepsia | | | |
| Abdominal pain lower | | | |
| Oral discomfort | | | |
| Mouth ulceration | | | |
| Lip swelling | | | |
| Psychiatric disorders | | | |
| Suicidal ideation | | | |
| Insomnia | | | |
| Anxiety | | | |
| Depression | | | |
| Depressed mood | | | |
| Suicide attempt | | | |
| Self injurious behavior | | | |
| Panic attack | | | |
| Depression suicidal | | | |
| Delirium | | | |
| Anhedonia | | | |
| Alcohol withdrawal syndrome | | | |
| Agitation | | | |
| Restlessness | | | |
| Psychotic disorder | | | |
| Paranoia | | | |

| System Organ Class/<br>Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Mania | | | |
| Loss of libido | | | |
| Hypomania | | | |
| Affective disorder | | | |
| Drug abuse | | | |
| Nervous system disorders | | | |
| Headache | | | |
| Somnolence | | | |
| Syncope | | | |
| Migraine | | | |
| Dizziness | | | |
| Seizure | | | |
| Carpal tunnel syndrome | | | |
| Tremor | | | |
| Restless legs syndrome | | | |
| Paraesthesia | | | |
| Lethargy | | | |
| Hypoaesthesia | | | |
| Formication | | | |
| Facial paresis | | | |
| Burning sensation | | | |
| Sedation | | | |
| Sciatica | | | |
| Ageusia | | | |
| Loss of consciousness | | | |
| Infections and infestations | | | |
| Bronchitis | | | |
| Upper respiratory tract infection | | | |
| Cellulitis | | | |
| Influenza | | | |
| Abscess limb | | | |
| Pneumonia | | | |
| Urinary tract infection | | | |
| Sinusitis | | | |
| Gastroenteritis | | | |
| Eye infection | | | |
| Bursitis infective | | | |

| System Organ Class/<br>Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Aspergilloma | . , | , , | |
| Acarodermatitis | | | |
| Tooth abscess | | | |
| Subcutaneous abscess | | | |
| Abscess neck | | | |
| Nasopharyngitis | | | |
| Muscle abscess | | | |
| Lung infection | | | |
| Kidney infection | | | |
| Injection site abscess | | | |
| Hepatitis viral | | | |
| Groin abscess | | | |
| Gingival abscess | | | |
| Gastroenteritis viral | | | |
| Injury, poisoning and procedural complications | | | |
| Overdose | | | |
| Laceration | | | |
| Contusion | | | |
| Limb injury | | | |
| Ligament sprain | | | |
| Eye contusion | | | |
| Muscle strain | | | |
| Joint injury | | | |
| Joint dislocation | | | |
| Head injury | | | |
| Tooth injury | | | |
| Tooth fracture | | | |
| Burns third degree | | | |
| Tendon injury | | | |
| Skin abrasion | | | |
| Road traffic accident | | | |
| Periorbital haematoma | | | |
| Nerve injury | | | |
| Multiple fractures | | | |
| Lower limb fracture | | | |
| Avulsion fracture | | | |
| Limb crushing injury | | | |

| System Organ Class/ Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Musculoskeletal and connective tissue disorders | | , | |
| Back pain | | | |
| Arthralgia | | | |
| Myalgia | | | |
| Joint swelling | | | |
| Neck pain | | | |
| Musculoskeletal pain | | | |
| Pain in extremity | | | |
| Muscle contracture | | | |
| Arthritis | | | |
| Temporomandibular joint syndrome | | | |
| General disorders and administration site conditions | | | |
| Chest pain | | | |
| Peripheral swelling | | | |
| Oedema peripheral | | | |
| Fatigue | | | |
| Drug withdrawal syndrome | | | |
| Chills | | | |
| Asthenia | | | |
| Pyrexia | | | |
| Pain | | | |
| Local swelling | | | |
| Feeling jittery | | | |
| Investigations | | | |
| Transaminases increased | | | |
| Hepatic enzyme increased | | | |
| White blood cell count decreased | | | |
| Liver function test increased | | | |
| Blood urine present | | | |
| Skin and subcutaneous tissue disorders | | | |
| Hyperhidrosis | | | |
| Rash | | | |
| Pruritus | | | |
| Urticaria | | | |
| Ecchymosis | | | |
| Cold sweat | | | |
| Alopecia | | | |

| System Organ Class/ Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Respiratory, thoracic and mediastinal disorders | . , | , | . , |
| Oropharyngeal pain | | | |
| Cough | | | |
| Rhinorrhoea | | | |
| Epistaxis | | | |
| Throat tightness | | | |
| Sinus congestion | | | |
| Respiratory depression | | | |
| Nasal congestion | | | |
| Asthma | | | |
| Eye disorders | | | |
| Vision blurred | | | |
| Eye irritation | | | |
| Dry eye | | | |
| Diplopia | | | |
| Amaurosis fugax | | | |
| Metabolism and nutrition disorders | | | |
| Decreased appetite | | | |
| Dehydration | | | |
| Hyponatraemia | | | |
| Hypokalaemia | | | |
| Gout | | | |
| Vascular disorders | | | |
| Hot flush | | | |
| Hypertension | | | |
| Renal and urinary disorders | | | |
| Nephrolithiasis | | | |
| Urinary retention | | | |
| Pollakiuria | | | |
| Haematuria | | | |
| Dysuria | | | |

| Table 35: Summary of Treatment Emergent* MedDRA Coded Adverse Events by Treatment Arm | | | |
|---|---|---|---|
| System Organ Class/<br>Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Reproductive system and breast disorders | | | |
| Vaginal discharge | | | |
| Menstruation delayed | | | |
| Breast mass | | | |
| Breast discharge | | | |
| Hepatobiliary disorders | | | |
| Hepatic failure | | | |
| Cholecystitis | | | |
| Surgical and medical procedures | | | |
| Tooth extraction | | | |
| Cardiac disorders | | | |
| Tachycardia | | | |
| Social circumstances | | | |
| Victim of crime | | | |
| Product issues | | | |
| Device deployment issue | | | |
| Pregnancy, puerperium and perinatal conditions | | | |
| Ectopic pregnancy | | | |

<sup>\*</sup>Note: treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.

| System Organ Class/ Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Participants with at least one treatment emergent serious adverse event | | , | . , |
| Psychiatric disorders | | | |
| Suicidal ideation | | | |
| Suicide attempt | | | |
| Self injurious behavior | | | |
| Psychotic disorder | | | |
| Depression suicidal | | | |
| Depression | | | |
| Delirium | | | |
| Anxiety | | | |
| Affective disorder | | | |
| Injury, poisoning and procedural complications | | | |
| Overdose | | | |
| Multiple fractures | | | |
| Burns third degree | | | |
| Infections and infestations | | | |
| Cellulitis | | | |
| Abscess limb | | | |
| Pneumonia | | | |
| Influenza | | | |
| Groin abscess | | | |
| Gastroenteritis | | | |
| Bronchitis | | | |
| Nervous system disorders | | | |
| Syncope | | | |
| Seizure | | | |
| Facial paresis | | | |
| Respiratory, thoracic and mediastinal disorders | | | |
| Respiratory depression | | | |
| Asthma | | | |
| Musculoskeletal and connective tissue disorders | | | |
| Back pain | | | |
| Metabolism and nutrition disorders | | | |
| Dehydration | | | |
| Hepatobiliary disorders | | | |
| Hepatic failure | | | |

| Table 36: Summary of Treatment Emergent* MedDRA Coded Serious Adverse Events by Treatment Arm | | | |
|---|---|---|---|
| System Organ Class/<br>Preferred Term (MedDRA v19.0 or higher) | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| General disorders and administration site conditions | | | |
| Chest pain | | | |
| Gastrointestinal disorders | | | |
| Vomiting | | | |
| Eye disorders | | | |
| Diplopia | | | |
| Pregnancy, puerperium and perinatal conditions | | | |
| Ectopic pregnancy | | | |

<sup>\*</sup>Note: treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.

CTN-0051: X:BOT
Statistical Analysis Plan

Version 3.0
April 27, 2017

# Table 37: Listing of Treatment Emergent\* Adverse Events by Treatment Arm [Serious Adverse Events Noted in Grey] Treatment Arm = BUP-NX

| | | | | | | | | | MedDRA | |
|---|---|---|---|---|---|---|---|---|---|---|
| СТР | Participant<br>ID | AE<br>Description | Onset<br>date | Severity<br>of AE | Relatedness | Outcome | Resolution<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ Class |

<sup>\*</sup>Note: treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.

CTN-0051: X:BOT
Statistical Analysis Plan

Version 3.0
April 27, 2017

Table 38: Listing of Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm

[Serious Adverse Events Noted in Grey]

Treatment Arm = BUP-NX

| | | | | | | | | MedDRA | | |
|---|---|---|---|---|---|---|---|---|---|---|
| СТР | Participant<br>ID | AE<br>Description | Onset<br>date | Severity<br>of AE | Relatedness | Outcome | Resolution<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ Class |

<sup>\*</sup>Note: treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.

CTN-0051: X:BOT
Statistical Analysis Plan

Version 3.0
April 27, 2017

Table 38: Listing of Non-Treatment Emergent Adverse Events in Randomized Participants by Treatment Arm

[Serious Adverse Events Noted in Grey]

Treatment Arm = XR-NTX

| | | | | | | | | | Me | dDRA |
|---|---|---|---|---|---|---|---|---|---|---|
| СТР | Participant<br>ID | AE<br>Description | Onset<br>date | Severity<br>of AE | Relatedness | Outcome | Resolution<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ Class |

<sup>\*</sup>Note: treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.

| Table 39: Listing of Non-Treatment Emergent Adverse Events Among Screen Failures [Serious Adverse Events noted in Grey] | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| СТР | Participant<br>ID | AE<br>Description | Onset date | Severity<br>of AE | Relatedness | Outcome | Resolution<br>Date | AE<br>Associated<br>With | Preferred<br>Term | System<br>Organ Class |

#### **SAE Narratives**

| | Table 40: Listing of Serious Adverse Events by Treatment Arm |
|---|---|
| Treatment Arm = BUP-NX | |
| | MedDRA |
| СТР | Participant AE Onset Severity CTP ID Description date of AE Relatedness Outcome Date AE AE Associated Preferred System Organ Class |

Note: MedDRA v19.0 or higher.

| | Table 40: Listing of Serious Adverse Events by Treatment Arm Treatment Arm = XR-NTX |
|---|---|
| | MedDRA |
| СТР | Participant AE Onset Severity CTP ID Description date of AE Relatedness Outcome Date AE Associated Preferred Organ Clas |

| Table 41: Listing of Deaths by Treatment Arm | |
|---|---|
| Treatment Arm=BUP-NX | |
| MedDRA | |
| СТР | CTP Participant AE Onset Relatedness Preferred System Organ Clas |

Note: MedDRA v19.0 or higher.

| Table 41: Listing of Deaths by Treatment Arm Treatment Arm=XR-NTX |
|---|
| MedDRA |
| CTP Participant AE Onset Relatedness Preferred System ID Description date Term Organ Class |

## Table 42 Listing of Participants with HAM-D and/or CHRT Assessment Question Responses Indicating Potential Suicidality by Treatment Arm

#### **Treatment Arm = BUP-NX**

| | | | | HAM-D Assessment | Cŀ | IRT Assessme | nt |
|---|---|---|---|---|---|---|---|
| СТР | Participant ID | Date of<br>Assessment | Study Day | Suicide | I have been<br>having<br>thoughts of<br>killing<br>myself | I have<br>thoughts<br>about how I<br>might kill<br>myself | I have a<br>plan to kill<br>myself |
| OV Maryhaven | | | | | | | |
| FL Gateway Community Services | | | | | | | |
| PA Tarzana Treatment Centers | | | | | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | | | | | | | |
| GNY Bellevue Hospital Center | | | | | | | |
| PNW ETS/RCKC | | | | | | | |
| MA Avery Road | | | | | | | |
| SW Turquoise Lodge Hospital | | | | | | | |
| OV Maryhaven | | | | | | | |
| FL Gateway Community Services | | | | | | | |
| PA Tarzana Treatment Centers | | | | | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | | | | | | | |
| GNY Bellevue Hospital Center | | | | | | | |
| PNW ETS/RCKC | | | | | | | |
| MA Avery Road | | | | | | | |
| SW Turquoise Lodge Hospital | | | | | | | |

Refer to figures for details regarding the color-coding.

### Table 42 Listing of Participants with HAM-D and/or CHRT Assessment Question Responses Indicating Potential Suicidality by Treatment Arm

#### **Treatment Arm = XR-NTX**

| | | | | HAM-D Assessment | CH | IRT Assessme | nt |
|---|---|---|---|---|---|---|---|
| СТР | Participant ID | Date of<br>Assessment | Study Day | Suicide | I have been<br>having<br>thoughts of<br>killing<br>myself | I have<br>thoughts<br>about how I<br>might kill<br>myself | I have a<br>plan to kill<br>myself |
| OV Maryhaven | | | | | | | |
| FL Gateway Community Services | | | | | | | |
| PA Tarzana Treatment Centers | | | | | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | | | | | | | |
| GNY Bellevue Hospital Center | | | | | | | |
| PNW ETS/RCKC | | | | | | | |
| MA Avery Road | | | | | | | |
| SW Turquoise Lodge Hospital | | | | | | | |
| OV Maryhaven | | | | | | | |
| FL Gateway Community Services | | | | | | | |
| PA Tarzana Treatment Centers | | | | | | | |
| NEC Stanley Street Treatment and Resources (SSTAR) | | | | | | | |
| GNY Bellevue Hospital Center | | | | | | | |
| PNW ETS/RCKC | | | | | | | |
| MA Avery Road | | | | | | | |
| SW Turquoise Lodge Hospital | | | | | | | |

Refer to figures for details regarding the color-coding.

| Table 43: Summary of Participants with Reponses Indicate Treatment Arm | Table 43: Summary of Participants with Reponses Indicating Potential Suicidality by Treatment Arm | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Number of Participants who endorsed suicidal ideation on CHRT at Screening | | | |
| Number of Participants who endorsed suicidal ideation on CHRT at any Follow-up Visit | | | |
| Number of Participants who endorsed suicidal ideation <sup>1</sup> on HAM-D <sup>1</sup> at Screening | | | |
| Number of Participants who endorsed suicidal ideation on HAM-D at any Follow-up Visit | | | |
| Number of Participants who ever endorsed a suicide attempt <sup>2</sup> on the HAM-D at any Follow-up Visit | | | |
| Number of Participants with AE's MedDRA-coded as either Suicide attempt, Suicidal Ideation, Self injurious behavior or Depression suicidal | | | |

 $<sup>^{\</sup>rm 1}$  Indicated as a response of 1 or higher to the HAM-D Suicide Question.  $^{\rm 2}$  Indicated as a response of 4 on the HAM-D Suicide Question

Figure 18: Participant-level Plot of HAM-D Question 3: Suicide by Treatment Arm
Figure 18A: Treatment Arm = BUP-NX





Figure 18B: Treatment Arm = XR-NTX

Figure 19: Participant-level Plot of CHRT Question 14: I have been having thoughts of killing myself, by Treatment Arm

Figure 19A: Treatment Arm = BUP-NX





Figure 19B: Treatment Arm = XR-NTX

Figure 20: Participant-level Plot of CHRT Question 15: I have been having thoughts of how I might kill myself, by Treatment Arm

Figure 20A: Treatment Arm = BUP-NX





Figure 20B: Treatment Arm = XR-NTX

Figure 21: Participant-level Plot of CHRT Question 16: I have a plan to kill myself, by Treatment Arm

Figure 12A: Treatment Arm = BUP-NX





Figure 12B: Treatment Arm = XR-NTX

Figure 22: Participant-level Trajectories for Participants with Aspartate Aminotransferase > 225 IU/L by Treatment Arm



Example figure provided.

Figure 23: Participant-level Trajectories for Participants with Alanine Aminotransferase > 225 IU/L by Treatment Arm



Example figure provided.

| Та | Table 44: Listing of Liver Function Tests for ALT and AST exceeding 45 IU/L by Treatment Arm | | | |
|---|---|---|---|---|
| Treatment Arm=BUP-NX | | | | |
| Baseline Aspartate Aspartate Aminotransferase CTP Participant ID Aspartate Aminotransferase (IU/L) Baseline Aspartate Aminotransferase (IU/L) Follow-up Aspartate Aminotransferase (IU/L) (IU/L) Follow-up Aspartate Aminotransferase (IU/L) | | | | |
| | | Tr | eatmei | nt Arm=XR-NTX |
| Baseline Aspartate Aminotransferase CTP Baseline Aspartate Aminotransferase (IU/L) Baseline Aspartate Aminotransferase (IU/L) Baseline Alanine Aminotransferase (IU/L) Follow-up Aspartate Aminotransferase (IU/L) | | | | |

Yellow highlighted cells indicate liver function test results greater than 45 IU/L. Red highlighted cells indicate liver function tests results greater than 225 IU/L.

| Table 45: Summary of Injection Site Abnormalities by CTP | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | OV<br>Maryhaven | FL Gateway<br>Community<br>Services | PA Tarzana<br>Treatment<br>Centers | NEC Stanley<br>Street<br>Treatment and<br>Resources<br>(SSTAR) | GNY<br>Bellevue<br>Hospital<br>Center | PNW ETS/<br>RCKC | MA<br>Avery<br>Road | SW<br>Turquoise<br>Lodge<br>Hospital | Total |
| Number of Participants<br>Randomized to XR-NTX | | | | | | | | | |
| Number of Participants with<br>Injection Site Abnormality | | | | | | | | | |
| Number of Injection Site<br>Abnormalities Reported | | | | | | | | | |
| Type of Injection Site<br>Abnormality | | | | | | | | | |
| Pain | | | | | | | | | |
| Abscess | | | | | | | | | |
| Sterile abscess | | | | | | | | | |
| Necrosis | | | | | | | | | |
| Cellulitis | | | | | | | | | |
| Tenderness | | | | | | | | | |
| Induration | | | | | | | | | |
| Swelling | | | | | | | | | |
| Erythema (redness) | | | | | | | | | |
| Bruising | | | | | | | | | |
| Pruritus | | | | | | | | | |
| Nodule | | | | | | | | | |
| Hematoma | | | | | | | | | |
| Other | | | | | | | | | |
| Severity of Injection Site<br>Abnormality | | | | | | | | | |
| Mild | | | | | | | | | |
| Moderate | | | | | | | | | |
| Severe | | | | | | | | | |

**Table 46: Listing of Injection Site Abnormalities** 

| СТР | Participant ID | Date of<br>Injection | Injection<br>Number | Event<br>Start<br>Date | Event<br>Resolution<br>Date | Abnormal Event | Severity | Treatment |
|---|---|---|---|---|---|---|---|---|

Appropriately qualified and trained medical personnel examine the injection site on the next Medical Management visit following the Vivitrol administration.

| | Treatment Arm | |
|---|---|---|
| SOWS Composite Score | BUP-NX<br>(N=) | XR-NTX<br>(N=) |
| SOWS Composite Score Before Induction | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min | | |
| Max | | |
| SOWS Composite Score after Naloxone Challenge | | |
| N | N/A | |
| Mean | N/A | |
| SD | N/A | |
| Median | N/A | |
| Min | N/A | |
| Max | N/A | |
| SOWS Composite Score After Induction | | |
| N | | |
| Mean | | |
| SD | | |
| Median | | |
| Min | | |
| Max | | |
| Change in SOWS Composite Score between post<br>Naloxone Challenge SOWS and after induction SOWS | | |
| N | N/A | |
| Mean | N/A | |
| SD | N/A | |
| Median | N/A | |
| Min | N/A | |
| Max | N/A | |
| Change in SOWS Composite Score* | | |
| N | | |
| Mean | | |
| SD | | |

| Table 47: Summary of Withdrawal Symptoms (SOWS Composite Score) at Induction by Treatment Arm | | |
|---|---|---|
| | Treatme | Treatment Arm |
| SOWS Composite Score | BUP-NX<br>(N=) | XR-NTX<br>(N=) |
| Median | | |
| Min | | |
| Max | | |

At the induction visit for the XR-NTX group, the SOWS is administered three times, the first time within the hour prior to the naloxone challenge, the second time 10-30 minutes following the naloxone challenge, and the third time 1-3 times following the XR-NTX injection. At the induction visit for the BUP-NX group, the SOWS is administered twice, the first time within the hour prior to the BUP-NX dosing and the second time 1-3 hours following dosing.

The SOWS is a 16-item questionnaire with a maximal score of 4 per item (0=absent, 4=extremely) for a maximal composite score of 64.

\*Change in SOWS Composite Score is calculated as the SOWS Composite Score after induction minus the SOWS Composite Score before induction. Thus, a negative value indicates symptoms improvement whereas a positive value indicates worsening.

| Table 48: Listing of Pregnancies by Treatment Arm Treatment Arm=BUP-NX | | | | | | |
|---|---|---|---|---|---|---|
| СТР | Participant ID | Date of Randomization | Date Staff<br>Aware | Action Taken with<br>Study Drug | Pregnancy<br>Outcome | Date of<br>Pregnancy<br>Outcome |

| Table 48: Listing of Pregnancies by Treatment Arm | | | | | | |
|---|---|---|---|---|---|---|
| Treatment Arm=XR-NTX | | | | | | |
| СТР | Participant ID | Date of Randomization | Date Staff<br>Aware | Action Taken with<br>Study Drug | Pregnancy<br>Outcome | Date of<br>Pregnancy<br>Outcome |
#### **Live Birth Narratives**

| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
|---|---|---|---|
| Number of randomized participants with protocol deviations | | | |
| Total number of protocol deviations | | | |
| Number of major protocol deviations | | | |
| Type of major protocol deviation – N (%) | | | |
| Medication dosing errors (protocol specified dose not dispensed) | | | |
| Breach of Confidentiality | | | |
| Safety assessment (e.g. labs, ECG, clinical referral to care) not conducted per protocol | | | |
| Stratification error | | | |
| Unauthorized assessments and/or procedures conducted prior to obtaining informed consent | | | |
| Medication dispensed to ineligible participant | | | |
| Participant use of protocol prohibited medication | | | |
| Type of minor protocol deviation – N (%) | | | |
| Study assessments not completed/followed as per protocol | | | |
| Biologic specimen not collected/processed as per protocol | | | |
| AE/SAE reported out of protocol specified reporting timeframe | | | |
| Protocol required visit/assessment not scheduled or conducted | | | |
| Study medication management - Other | | | |
| Study procedures/assessments - Other | | | |
| AE not reported | | | |
| Laboratory assessments - Other | | | |
| Non IRB approved/outdated/obsolete informed consent documents used | | | |
| Informed consent process not properly conducted and/or documented | | | |
| Informed consent procedures - Other | | | |
| Invalid/incomplete informed consent form | | | |

| Table 49: Summary of Protocol Deviations in Randomized Participants, by<br>Treatment Arm | | | |
|---|---|---|---|
| | BUP-NX<br>(N=) | XR-NTX<br>(N=) | Total<br>(N=) |
| Adverse event - Other | | | |
| Other significant deviations | | | |
| Inclusion/exclusion criteria - Other | | | 1 |
| AE/SAE not elicited, observed and/or documented as per protocol | | | |
| Randomization procedures - Other | | | |
| Study behavioral intervention was not provided/performed as per protocol | | | |

| Table 50: Summary of Protocol Deviations Among So | reen Failures |
|---|---|
| | Total<br>(N=) |
| Number of screen failures | |
| Number of screen failures with protocol deviations | |
| Total number of protocol deviations | |
| Number of major protocol deviations | |
| Type of major protocol deviation – N (%) | |
| Participant use of protocol prohibited medication | |
| Breach of Confidentiality | |
| Type of minor protocol deviation – N (%) | |
| Non IRB approved/outdated/obsolete informed consent documents used | |
| Study assessments not completed/followed as per protocol | |
| Biologic specimen not collected/processed as per protocol | |
| Invalid/incomplete informed consent form | |
| Informed consent process not properly conducted and/or documented | |
| Other significant deviations | |

## Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category Deviation Category=Informed Consent Procedures

| СТР | Participant<br>ID | Treatment<br>Arm | Date of Deviation | Days from<br>Site<br>Endorsement | Date<br>Entered<br>in<br>AdvEDC | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|---|

## Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category Deviation Category=Laboratory Assessments

| СТР | Participant<br>ID | Treatment<br>Arm | Date of<br>Deviation | Days from<br>Site<br>Endorsement | Date<br>Entered<br>in<br>AdvEDC | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | · | | | | | |

## Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category Deviation Category=Study Procedures/assessments

| СТР | Participant<br>ID | Treatment<br>Arm | Date of<br>Deviation | Days from<br>Site<br>Endorsement | Date<br>Entered<br>in<br>AdvEDC | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|---|

# Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category Deviation Category=Adverse Event

| СТР | Participant<br>ID | Treatment<br>Arm | Date of Deviation | Days from<br>Site<br>Endorsement | in | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|---|

## Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category Deviation Category=Randomization Procedures

| СТР | Participant<br>ID | Treatme<br>nt Arm | Date of<br>Deviatio<br>n | Days from<br>Site<br>Endorsemen<br>t | Date<br>Entered<br>in<br>AdvED<br>C | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to<br>Prevent<br>Recurrence | IRB<br>Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|---|

## Table 51: Listing of Protocol Deviations in Randomized Participants by Deviation Category Deviation Category=Study Medication Management

| СТР | Participant<br>ID | Treatment<br>Arm | Date of<br>Deviation | Days from<br>Site<br>Endorsemen<br>t | Date<br>Entered<br>in<br>AdvEDC | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB<br>Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|---|

| | Table 52: Listing of Protocol Deviations among Screen Failures by Deviation Category | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Deviation Category=Informed Consent Procedures | | | | | | | | |
| СТР | Participant<br>ID | Date of<br>Deviation | Days from Site<br>Endorsement | Date Entered in AdvEDC | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB<br>Reporting<br>Required? |

# Table 52: Listing of Protocol Deviations Among Screen Failures by Deviation Category Deviation Category=Study Procedures/Assessments

| СТР | Participant<br>ID | Date of<br>Deviation | Days from<br>Site<br>Endorsement | Date Entered<br>in AdvEDC | Level<br>of<br>Deviation | Deviation<br>Type | Description | Plan to Prevent<br>Recurrence | IRB<br>Reporting<br>Required? |
|---|---|---|---|---|---|---|---|---|---|

| | Table 52: Listing of Protocol Deviations Among Screen Failures by Deviation Category Deviation Category=Other Significant Deviations | |
|---|---|---|
| Participant Date of Deviation Description Description Description Recurrence Required | | |
| | | - |